### The GlaxoSmithKline group of companies

200331

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A Phase I, Open-Label, Dose-Finding Study of GSK2636771 Administered in Combination with Enzalutamide (Xtandi) in Male Subjects with Metastatic Castration-Resistant Prostate Cancer (mCRPC) |
|---|---|---|
| <b>Compound Number</b> | : | GSK2636771 |
| <b>Effective Date</b> | : | 03-MAR-2020 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2013N172718 04.
- This RAP is intended to describe the safety, efficacy and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author(s):**

| Author | Date |
|------------------------------------------------|-------------|
| Lead | |
| PPD | |
| Statistician (Oncology, Clinical Statistics) | |
| Co-Authors | |
| PPD | 17-FEB-2020 |
| Clinical Pharmacology Manager (Oncology, CPMS) | |
| PPD | 17 EED 2020 |
| Clinical Biomarker Lead (Oncology, Biomarkers) | 17-FEB-2020 |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

200331

## **RAP Team Review Confirmations (Method: E-mail)**

| Reviewer | Date |
|---------------------------------------------------------------|-------------|
| Clinical Development Director (Oncology) | 17-FEB-2020 |
| Principal Programmer/Analyst (Oncology, Clinical Programming) | 18-FEB-2020 |

# Clinical Statistics and Clinical Programming Line Approvals (Method: Pharma TMF eSignatures)

| Approver | Date |
|------------------------------------------------------------|-------------|
| Senior Statistics Director (Oncology, Clinical Statistics) | e-signature |
| Programming Manager (Oncology, Clinical Programming) | e-signature |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | | IONAmendments | |
| 2. | <ul><li>2.1. Change</li><li>2.2. Study</li><li>2.3. Study</li></ul> | OF KEY PROTOCOL INFORMATION ges to the Protocol Defined Statistical Analysis Plan Objective(s) and Endpoint(s) Design tical Hypotheses / Statistical Analyses | 8<br>8<br>11 |
| 3. | 3.1. Interin<br>3.1.1.<br>3.1.2. | | 13<br>13<br>13 |
| 4. | | OPULATIONS | |
| 5. | CONVENTIO<br>5.1. Study<br>5.2. Baseli<br>5.3. Other | TIONS FOR DATA ANALYSES AND DATA HANDLING NS Treatment & Sub-group Display Descriptors ine Definitions Considerations for Data Analyses and Data Handling | 16<br>16 |
| 6. | | Demographic and Baseline Characteristics Treatment Compliance | 18<br>18<br>19<br>19 |
| 7. | 7.2. Prima 7.2.1. 7.2.2. 7.2.3. | iew of Planned Efficacy Analyses ry Efficacy Analyses Endpoint / Variables | 21<br>22<br>24<br>25<br>25<br>27 |
| | 7.2.4. 7.3. Secon 7.3.1. 7.3.2. 7.3.3. | ndary Efficacy Analyses<br>Endpoint / Variables<br>Summary Measure | 28<br>28<br>32 |

| | | 7.3.4. | Statistical Analyses / Methods | 32 |
|---|---|---|---|---|
| 8. | SAFE | Γν ανιαι ν | /SES | 3/1 |
| 0. | 8.1. | | v of Planned Analyses | |
| | 8.2. | | f Exposure | |
| | 8.3. | | Events Analyses | |
| | 8.4. | | Events of Special Interest (AESI) Analyses | |
| | 8.5. | | _aboratory Analyses | |
| | 8.6. | | afety Analyses | |
| | 0.0. | 8.6.1. | Deaths and Serious Adverse Events | |
| | 8.7. | | cies | |
| ^ | | | IETIC ANALYCEC | 20 |
| 9. | | | NETIC ANALYSES | |
| | 9.1. | | Pharmacokinetic Analyses | |
| | 9.2. | | ary Pharmacokinetic Analyses | |
| | | 9.2.1. | Endpoint / Variables | |
| | | | 9.2.1.1. Drug Concentration Measures | |
| | | 9.2.2. | Population of Interest | |
| | | 9.2.3. | Statistical Analyses / Methods | 36 |
| 10. | BIOMA | ARKER A | NALYSES | 37 |
| | 10.1. | Explorate | ory Biomarker Analyses | 37 |
| | | 10.1.1. | | |
| | | | 10.1.1.1. Circulating Tumour Cells | |
| | | | 10.1.1.2. Frequency of PTEN loss and Mechanism of PTEN Loss | |
| | | | 10.1.1.3. Mutational Analysis of Tumour Biopsy Sample | |
| | | 10.1.2. | Summary Measure | |
| | | 10.1.2. | Population of Interest | |
| | | 10.1.4. | Statistical Analyses / Methods | |
| | | | • | |
| 11. | PHAR | MACOKIN | NETIC / PHARMACODYNAMIC ANALYSES | 39 |
| 12. | REFE | RENCES. | | 40 |
| 12 | ٨٥٥٢١ | NDICES | | 11 |
| 13. | 13.1. | | x 1: Protocol Deviation Management and Definitions for Per | 41 |
| | 13.1. | | Population | 11 |
| | | 13.1.1. | | |
| | 13.2. | | x 2: Schedule of Activities | 41<br>42 |
| | 13.2. | 13.2.1. | | 42 |
| | 13.3. | | x 3: Assessment Windows | |
| | 13.3. | 13.3.1. | | |
| | 12.4 | | | 50 |
| | 13.4. | | x 4: Study Phases and Treatment Emergent Adverse | 57 |
| | | 13.4.1. | , | |
| | 12 F | 13.4.2. | Treatment Emergent Flag for Adverse Events | |
| | 13.5. | | x 5: Data Display Standards & Handling Conventions | |
| | | 13.5.1. | Reporting Process | |
| | | 13.5.2. | Reporting Standards | |
| | 12.0 | 13.5.3. | Reporting Standards for Pharmacokinetic | |
| | 13.6. | Appendi | x 6: Derived and Transformed Data | 60 |

| | | | 200331 |
|---|---|---|---|
| | 13.6.1. | General | 60 |
| | 13.6.2. | Study Population | 61 |
| | 13.6.3. | Efficacy | 61 |
| | 13.6.4. | Safety | |
| 13.7. | Appendix | x 7: Reporting Standards for Missing Data | 64 |
| | 13.7.1. | | 64 |
| | 13.7.2. | 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 | |
| | | 13.7.2.1. Handling of Missing and Partial Dates | 64 |
| 13.8. | Appendix | x 8: Values of Potential Clinical Importance | 67 |
| | | Laboratory Values | |
| | | ECG and Vital Signs | |
| 13.9. | | x 9: Population Pharmacokinetic (PopPK) Analyses | |
| | | x 10: Pharmacokinetic / Pharmacodynamic Analyses | |
| 13.11. | | x 11: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 13.12. | | x 12: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | | Safety Figures | |
| | | Pharmacokinetic Tables | |
| | | .Pharmacokinetic Figures | |
| | | .Biomarker Tables | |
| | | Biomarker Figures | |
| | | ICH Listings | |
| | | Non-ICH Listings | |
| 13.13. | Appendix | x 13: Example Mock Shells for Data Displays | 100 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 200331:

| Revision Chronology: | | |
|---|---|---|
| 2013N172718_00 | 22-May-2014 | Original |
| 2013N172718_01 | 08-Sep-2014 | Amendment 1 incorporates changes to Section 5.2, Permanent Discontinuation of Study Treatment(s) for clarification as requested by the Medicines and Healthcare products Regulatory Agency (MHRA) in the United Kingdom. |
| 2013N172718_02 | 26-Feb-2015 | Amendment 2 incorporates changes to list of authors and primary medical monitor (contact information) due to changes in personnel assignment within GSK; list of abbreviations was revised appropriately based upon addition/deletion of abbreviated terms used throughout the protocol; Time and Events Tables were revised for clarification of assessments and procedures to be performed and to reflect changes made throughout the body of the protocol. |
| 2013N172718_03 | 24-Jun-2016 | Amendment 3 incorporates changes to update the risk assessment section and to include additional requirements for monitoring of renal events following an INDSR report for Acute Renal Failure in a subject enrolled in this study. In addition, it was clarified that subjects with disease progression defined by PSA progression alone or for the worsening of an isolated disease site that is not clinically significant are not required to discontinue treatment in the study. Separate definitions for disease progression as a study endpoint and disease progression mandated by the protocol to result in a subject being withdrawal from treatment is clarified. Optional pharmacodynamics paired biopsies as well as clarifications around biomarker assessments were added to the Time and Events tables for the Dose Escalation and Dose Expansion Phases. Additional language was added to clarify that the decision to terminate the Dose Expansion Phase will take into account all relevant factors, including but not solely based upon the statistical methodology and futility criterion. Other minor clarifications and corrections of inadvertent errors were also added. |
| 2013N172718_04 | 27-Jan-2017 | Amendment 4 was completed to include additional requirements for monitoring of events related to calcium results, including revisions to the Table & Events to clarify additional laboratory testing requirements; clarification of secondary clinical activity endpoints and update to associated statistical section(s); revision of clinical activity population allowing the combination of dose escalation and dose |

200331

| Revision Chronology: | |
|---|---|
| | expansion populations; revision of dose escalation and dose expansion wording to allow multiple dose levels in dose expansion to establish RP2D after dose expansion phase; adjustment to Week 12 visit window and clarification for Week 12 assessment timing; revision to reflect current indication for enzalutamide throughout; clarification of study populations; clarification of bone progression definition. |
| | Other minor clarifications and corrections of inadvertent errors were also added. |

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

## 1.1. RAP Amendments

Revision chronology:

| RAP Section Amendment Details | |
|---|---|
| Reporting and Analysis Plan_200331_Final_V1 [02-Dec-2019] | |
| Reporting and Analysis Pla | n_200331_Amendment_Final_V1 |
| 7.2. | Removed references to PCWG2 modification of RECIST since it was not required in the protocol. Removed the text "PCWG2 modified" prior to "RECIST" throughout the section. Removed the text "Additional requirement (per PCWG2) that progression at first assessment be confirmed by a second scan 6 or more weeks later" from the RECIST response (at 16 weeks) in Table 2. |
| 7.2.1.2. | Added the following text to Table 4 to clarify the definition of Bone Response (at week 12): "This algorithm assumes subjects had bone lesions identified via bone scan at baseline. For subjects without bone lesions identified via Bone Scan at baseline, the confirmed and unconfirmed bone responses are set to missing." |
| 7.2.1.3. | Removed the following text from the RECIST response as was not required in the protocol: "with the added PCWG2 requirement that progression at first assessment be confirmed by a second scan 6 or more weeks later." |
| 7.2.1.4. | Added additional 12 scenarios to Table 5 to clarify the Overall<br>Response at week 12. These scenarios take into account subjects with<br>no baseline bone lesions identified via bone scan. |
| 7.3.1. | Removed the text "PCWG2 modified" prior to "RECIST" throughout the section as was not required in the protocol. |
| 9.2.1.1. | Clarified the description of the how the secondary objectives will be displayed. |
| 13.12.9., 13.12.10.,<br>13.12.14. | Added clarifying text to the titles of the PK tables/figures/listings |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol amendment 4 (Dated: 27-Jan-2017) are outlined in Table 1. These exploratory endpoints were unlikely to provide any additional information to what would be provided by the other endpoints.

Table 1 Exploratory Endpoints Removed from Protocol Defined Analysis Plan

| Protocol | | Reporting & Analysis Plan | |
|---|---|---|---|
| objective | endpoint | Statistical Analysis<br>Plan | Rationale for Changes |
| Evaluation of<br>biomarkers in<br>CTCs that may<br>predict response<br>to combination | AR expression, PTEN FISH and other genomic evaluations in CTCs | • removed | analysis not performed since no response was identified |
| Evaluation of tumor tissue to explore explanation for the mechanism of resistance to combination therapy | Based on analysis of DNA, RNA and proteins from tumour tissue obtained at time of progression after initially responding to combination therapy | • removed | paired biopsies were not obtained |
| To determine pharmacodynamic effects of drug treatment | RNA/protein analysis of pre/post treatment tumour biopsies | • removed | paired biopsies were not obtained |

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| <ul> <li>To assess the safety and<br/>tolerability of GSK2636771 +<br/>enzalutamide administered<br/>orally once daily continuously in<br/>subjects with mCRPC.</li> </ul> | <ul> <li>AEs, SAEs, DLTs, and changes in laboratory<br/>values, ECGs, and vital signs (BP, temperature<br/>and heart rate)</li> </ul> |
| <ul> <li>To determine the RP2D of<br/>orally administered<br/>GSK2636771 + enzalutamide<br/>in subjects with mCRPC.</li> </ul> | <ul> <li>Safety and tolerability as assessed by AEs,<br/>SAEs, DLTs, and changes in laboratory values,<br/>ECGs, and vital signs (BP, temperature and<br/>heart rate)</li> </ul> |

200331

| Objectives | Endpoints |
|---|---|
| To evaluate lack of progression in the dose expansion subjects with mCRPC by rate of subjects who do not progress for 12 weeks | Non-Progressive Disease (Non-PD) rate for 12 weeks according to PCWG2 criteria (either by RECIST 1.1, or progression in bone or PSA progression with accompanying progression by RECIST 1.1 or bone scan when baseline radiological or bone disease present or PSA progression if no other baseline disease). |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the clinical activity of oral GSK2636771 + enzalutamide in the treatment of mCRPC (PTEN deficient) To determine the effect of | <ul> <li>PSA50 response rate defined as the percent of subjects achieving PSA50 at 12 weeks or thereafter (PSA50 is ≥50% decrease in PSA from baseline)</li> <li>Objective Response Rate (ORR) defined as complete response (CR) rate plus partial response (PR) rate per RECIST 1.1</li> <li>Time to PSA progression according to PCWG2 criteria</li> <li>Time to radiological progression according to PCWG2 criteria (either by RECIST 1.1, PSA progression and/or progression in bone)</li> <li>Radiological progression free survival (rPFS) per RECIST1.1 and/or bone scans</li> <li>Plasma concentrations of enzalutamide and</li> </ul> |
| GSK2636771 on enzalutamide PK following repeat-dose oral administration. | N-desmethyl enzalutamide. |
| <ul> <li>To determine the PK of<br/>GSK2636771 in the presence<br/>of enzalutamide.</li> </ul> | Blood GSK2636771 concentrations. |
| Exploratory Objectives | Exploratory Endpoints |
| To determine the frequency of<br>PTEN deficiency in subjects<br>with mCRPC | <ul> <li>Frequency of PTEN-deficient mCRPC reported<br/>in subjects based on pre-screened tumours</li> </ul> |
| To determine the mechanism of<br>PTEN deficiency | <ul> <li>PTEN deletion, mutation or promoter<br/>methylation</li> </ul> |
| <ul> <li>To identify additional<br/>biomarkers (DNA, RNA or<br/>protein based) in tumour or in<br/>circulation that may predict<br/>response to oral GSK2636771<br/>+ enzalutamide</li> </ul> | <ul> <li>Response prediction biomarkers based on<br/>analysis of DNA, RNA, and proteins from<br/>surrogate tissues (e.g., cfDNA) and/or tumour<br/>tissue</li> </ul> |
| To determine the effect of<br>enzalutamide with<br>GSK2636771 on the kinetics of<br>tumour growth | Longitudinal tumour size measurements; serum PSA levels, change from baseline in CTCs |

200331

| Objectives | Endpoints |
|---|---|
| <ul> <li>Evaluation of biomarkers in<br/>CTCs that may predict<br/>response to combination</li> </ul> | AR expression, PTEN FISH and other genomic evaluations in CTCs |
| <ul> <li>Evaluation of tumour tissue to<br/>explore explanation for the<br/>mechanism of resistance to<br/>combination therapy</li> </ul> | Based on analysis of DNA, RNA and proteins<br>from tumour tissue obtained at time of<br>progression after initially responding to<br>combination therapy |
| To determine pharmacodynamic effects of drug treatment | RNA/protein analysis of pre/post treatment tumour biopsies |

## 2.3. Study Design

| Overview of S | Study Desig | n and Key I | Features | |
|---|---|---|---|---|
| Design<br>Features | Dose Escalation Phase of the study is to determine the maximum tolerated dose (MTD) and select a recommended dose for Dose Expansion Phase or a recommended Phase 2 dose (RP2D) based on the safety, pharmacokinetic, and pharmacodynamic profiles observed after combination therapy of GSK2636771 and enzalutamide. Any cohort may be expanded up to 12 subjects in order to collect adequate data on safety, PD or PK. | | | |
| | Dose Expansion Phase: This phase of the study will evaluate the long-term safety of the combination treatment as well as the 12-week non-progressive disease (PD) rate of the combination treatment in subjects with mCPRC. To confirm dose(s) identified during dose escalation, multiple dose levels of GSK2636771 in combination with enzalutamide may be examined during dose expansion, with each dose level cohort enrolling up to 20 subjects. | | | |
| Dosing | The planned starting dose of study treatment will be GSK2636771 300 mg orally once daily in combination with enzalutamide 160 mg orally once daily. Participants will begin combination therapy only after completing a 14-day run-in period of enzalutamide monotherapy 160 mg orally once daily. Dose escalations will be performed in Dose Escalation Phase and dose adjustments are allowed to address tolerability and safety issues. | | | |
| | Cohort | N | GSK2636771 | Enzalutamide |
| | -1 | 3 - 6 | 200 mg once daily | 160 mg once daily |
| | 1 | 3 - 6 | 300 mg once daily | 160 mg once daily |
| | 2 | 3 - 6 | 400 mg once daily | 160 mg once daily |
| Treatment | This is a non-randomized open-label study. | | | |
| Assignment | | | inalyses will be performed | |

200331

## 2.4. Statistical Hypotheses / Statistical Analyses

No formal statistical hypothesis will be tested during dose escalation phase. All analyses will be descriptive and exploratory.

For dose expansion phase, the 12-week non-PD rate will be tested using the predictive probability design by Lee and Liu (Lee, 2008). The null and alternative hypotheses for the non-PD rate are as follows:

H0: p≤ 5.0% HA: p>30%.

This hypothesis will be tested using a combination of data provided in both the dose escalation and dose expansion phases.

#### 3. PLANNED ANALYSES

### 3.1. Interim Analyses

#### 3.1.1. Dose Escalation Phase

In the Dose Escalation Phase, available safety data will be reviewed and summarized on an ongoing basis. Review of preliminary safety data from all available dose cohorts will be performed in each study treatment combination before starting a new dose cohort and before selecting a dose level for expansion. Safety will be reviewed on an ongoing basis by the Safety Monitoring Team, composed of study investigators and key GSK personnel including the medical monitor, study manager, and study statistician.

#### 3.1.2. Dose Expansion Phase

After the initial 10 subjects become evaluable at a dose level using a combination of dose escalation and dose expansion subjects, 12-week non-PD rate will be reviewed on an ongoing basis and the number of responses observed will be compared with the stopping rules provided below.

## 3.2. Final Analyses

The final planned primary and secondary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed or withdrawn from the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

200331

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screened | This population will consist of all subjects who were screened for PTEN status and enrolment of study | <ul> <li>Summary of study<br/>eligibility and PTEN<br/>status</li> </ul> |
| All Treated Safety | <ul> <li>This population will consist of all subjects who<br/>receive at least one dose of GSK2636771 or<br/>Enzalutamide.</li> </ul> | Safety |
| All Treated<br>Clinical Activity | This population will consist of all subjects who received at least one dose of GSK2636771. | Clinical Activity |
| Modified All<br>Treated Clinical<br>Activity | This population will consist of all subjects in All Treated Clinical Activity who were treated at the same dose as the dose expansion cohort and have been on study drug for at least 12 weeks or have discontinued study treatment due to disease progression, died, or withdrawn for any reason. | Evaluation of non-<br>PD rate |
| All Evaluable<br>Subjects | This population will consist of all subjects from<br>All Treated Clinical Activity Population who<br>have at least one post-dose disease<br>assessment and have been exposed to study<br>drug for at least 12 weeks or have progressed<br>or have died or have withdrawn from the study<br>for any reason | Dose Escalation &<br>Expansion futility<br>analyses |
| PK Concentration<br>Population | This population will consist of all subjects in<br>the All Treated Safety Population for whom a<br>blood sample for pharmacokinetics is obtained,<br>analysed, and was measurable. | Listing, summary,<br>and figures of PK<br>concentration |
| Biomarker<br>Population | This population will consist of subjects in the All Treated Safety Population for whom a | PTEN deletion and gene mutation |
| | sample was obtained and analyzed for biomarkers | CTC conversion |

### NOTES:

 Please refer to Appendix 12: List of Data Displays which details the population to be used for each display being generated.

## 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

200331

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

Participants will be listed and summarized based on their treatment group initially assigned regardless of any dose modifications that may occur following treatment initiation.

| Treatment Group Descriptions | | | | |
|---|---|---|---|---|
| Ra | ndAll NG | Data Displa | | |
| Code | Description | Description | Data Display | Order in TLF |
| Α | Enzalutamide | Run-in Enzalutamide | Run-in Enza | 1 |
| | | GSK2636771 200mg/<br>Enzalutamide 160mg<br>Escalation | GSK 200mg / Enza 160mg<br>Escalation | 2 |
| | | GSK2636771 200mg/<br>Enzalutamide 160mg<br>Expansion | GSK 200mg / Enza 160mg<br>Expansion | 3 |
| В | GSK2636771 +<br>Enzalutamide | GSK2636771 200mg/<br>Enzalutamide 160mg<br>Overall | GSK 200mg / Enza 160mg<br>Overall | 4 |
| | | GSK2636771 300mg/<br>Enzalutamide 160mg<br>Escalation | GSK 300mg / Enza 160mg<br>Escalation | 5 |
| | | GSK2636771 400mg/<br>Enzalutamide 160mg<br>Escalation | GSK 400mg / Enza 160mg<br>Escalation | 6 |

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest GSK2636771 pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first GSK2636771 dose and used as baseline.

For laboratory data, baseline will be the latest non-missing pre-dose value from central lab. If no central lab value is available, the latest non-missing pre-dose value from local lab will be used. If there are multiple assessments on the same day, the mean will be used as the baseline value.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

200331

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 13.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 13.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 13.6 | Appendix 6: Derived and Transformed Data |
| 13.7 | Appendix 7: Reporting Standards for Missing Data |
| 13.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the All Treated Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, demographic and baseline characteristics, protocol deviations, substance use, past and current medical conditions, disease characteristics at initial diagnosis and at screening, prior and follow-up anti-cancer therapy, cancer-related surgical procedures, concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 12: List of Data Displays.

#### 6.1.1. Disposition of Subjects

A summary of the number of subjects in each of the dosing groups/phases will be provided. A listing of subjects excluded from analysis populations will also be provided.

A summary of subject status and reason for study withdrawal will be provided. This display will show the number and percentage of subjects who withdrew from the study, including primary reasons for study withdrawal. Reasons for study withdrawal will be presented in the order they are displayed in the eCRF.

A summary of study treatment status will be provided. This display will show the number and percentage of subjects who are completed or discontinued study treatment and a summary of the primary reasons for discontinuation of study treatment. Reasons for study treatment discontinuation will be presented in the order they are displayed in the eCRF. A listing of study treatment discontinuation will be generated. The listing will include last dose date and reasons for study treatment discontinuation as well as study part of discontinuation

A table of study eligibility information will be provided based on All Pre-screened and Screened population. Number of subjects who were pre-screened for PTEN status and/or screened for enrolment, reasons of failure, subjects PTEN status etc. will be presented.

#### 6.1.2. Demographic and Baseline Characteristics

The demographic characteristics (e.g. age, race, ethnicity, sex, baseline height, and baseline body weight) will be summarized and listed. In addition, age will also be categorized and summarized by two groups of categories, <18, 18-64, 65-74, >74 and <18-64, 65-84; >=85 for Development Safety Update Report and Europe Clinical Trial Registry disclosure, respectively. The count and percentage will be computed for sex and ethnicity.

Race and racial combinations will be summarized and listed.

Medical conditions will be summarized by past and current categories.

200331

Disease history and characteristics (primary tumor type, lesion status, time since initial diagnosis in weeks, stage at initial diagnosis and screening, time since last progression in weeks) will be listed. Separate summaries of disease characteristics at initial diagnosis and screening will be provided.

Prior anti-cancer therapy will be coded using GSK Drug coding dictionary, then summarized by type of therapy and listed. A listing of prior anti-cancer therapy will show the relationship between Anatomical Therapeutic Chemical (ATC) Level 1, Ingredient, and verbatim text.

A summary of prior anti-cancer therapies will be provided. The number of lines of prior anti-cancer therapies and radiotherapy will be tabulated. Number of subjects who received Enzalutamide before or after chemotherapy will be provided. Summary of cancer-related surgeries will be produced. A summary of the best response to the most recent prior anti-cancer therapy will also be provided.

Substance use, including smoking history and alcohol use, will also be summarized and listed.

#### 6.1.3. Treatment Compliance

A listing of planned and actual treatments will be produced including number of tablets prescribed per day and total number of tablets dispensed.

In addition, summaries of study treatment exposure by Enzalutamide run in and combination treatment with GSK2636771 and dose modifications (e.g. number of dose reductions, number of dose interruptions) will further characterize compliance.

#### 6.1.4. Concomitant Medications

Concomitant medications will be coded using GSK Drug coding dictionary, summarized, and listed. The summary of concomitant medications will show the number and percentage of subjects taking concomitant medications by Ingredient. Multi-ingredient products will be summarized by their separate ingredients rather than as a combination of ingredients.

In the summary of concomitant medications, each subject is counted once within each unique ingredient. For example, if a subject takes Amoxycillin on two separate occasions, the subject is counted only once under the ingredient "Amoxycillin". In the summary of concomitant medications, the ingredients will be summarized by the base only, using CMBASECD and CMBASE.

A summary of the relationship between concomitant medications and reasons of the medications will be generated.

Blood products or blood supportive care products will be listed.

200331

#### 6.1.5. Subsequent Anti-Cancer Therapies

The number and percentage of subjects that received chemotherapy, immunotherapy, hormonal therapy, biologic therapy, radioactive therapy, small molecule targeted therapy, radiotherapy and cancer-specific surgery as post study treatment (see Section 13.4.1 for definition) anti-cancer therapy will be summarized. Time from study treatment discontinuation to the first post study anti-cancer therapy will also be included in this summary table.

Follow-up anti-cancer therapy will be coded using GSK Drug coding dictionary, then summarized by ingredient. A listing of the type of follow-up anti-cancer therapy received (chemotherapy, immunotherapy, hormonal therapy, biologic therapy, radioactive therapy, small molecule targeted therapy, radiotherapy and cancer-specific surgery and details of the anticancer therapy for each subject will be provided.

#### 7. EFFICACY ANALYSES

## 7.1. Overview of Planned Efficacy Analyses

The primary efficacy analyses will be based on the All Treated Clinical Activity Population, unless otherwise specified, and all summaries and data listings will use treatment labels as specified in Section 5.1. All summaries will be presented by dose, and overall.

## 7.2. Primary Efficacy Analyses

This analysis is to determine whether the 12-week non-PD rate is greater than 5%. The 12-week non-PD rate is defined as the percentage of subjects without progression (non-PD) at Week 12 as determined from PSA results, radiographic assessment per RECIST 1.1, and bone scan (see Section 7.2.1.4 for algorithm details). The PSA and bone scan results recorded at week 12 will be used for the evaluation of 12-week non-PD rate. Radiological assessments (CT/MRI) of target and non-target lesions at week 16 (instead of week 12) will be considered for the evaluation of week 12 non-PD rate since there were no week 12 radiological assessments scheduled for subjects during the study.

The disease progression is defined by 1 or more of the following criteria:

- PSA progression alone if no other baseline disease
- PSA progression according to the PCWG2 criteria with accompanying progression by RECIST 1.1 or bone scan for subjects with soft tissue baseline disease
- Bone progression on bone scan according to the PCWG2 criteria [measured by bone scan]
- Radiographic progression in soft tissue or bone by RECIST 1.1 for subjects with baseline disease.

The components of the 12 week non-PD rate primary efficacy endpoint are defined in Table 2. Additional details on these endpoints and composite 12-week non-PD rate are provided in Section 7.2.1 through Section 7.2.4.

200331

Table 2 Components of the 12 week Non-PD Rate

| Primary Efficacy endpoint | Definition |
|---|---|
| PSA Response (at 12 weeks) | Progression Definition (per PCWG2)*: |
| | If there has been a decline from baseline: time from start of therapy to first PSA increase that is ≥25% and ≥2 ng/mL in absolute value from the nadir, and which is confirmed by a second value 3 or more weeks later (i.e., a confirmed rising trend) at least 12 weeks after the start of combination treatment |
| | If there has NOT been a decline from baseline: time from start of therapy to first PSA increase that is ≥25% and ≥2 ng/mL in absolute value from the baseline value, determined at least 12 weeks after start of combination treatment |
| | See Section 7.2.1 for additional details on response |
| Bone Response (at 12 weeks) | Progression Definition (per PCWG2)*: |
| | The appearance of ≥2 new lesions, and, for the first reassessment only, a confirmatory bone scan performed 6 or more weeks later that shows a minimum of 2 or more additional new lesions. The date of progression is the date of the first scan that shows a minimum of 2 additional new lesions. |
| | See Section 7.2.2 for additional details on response. |
| RECIST Response (at 16 | Progression Definition (per RECIST v1.1)*: |
| weeks) | At least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. The date of PD is the date of the first scan that shows progression. Progression is also defined as unequivocal progression in non-target lesions or identification of unequivocal new lesions. |
| | See Section 7.2.3 for additional details on response. |

<sup>\*[</sup>Scher, 2008]

## 7.2.1. Endpoint / Variables

## **7.2.1.1. PSA Response (at week 12)**

Determination of PSA response at week 12 is based on PCWG2 criteria. The algorithm is outlined in the Table 3. The response is categorized into progression (PD), non-PD, or not evaluable (NE).

200331

Table 3 Assessment of PSA Response

| Week 8 (or any<br>visit < 12 weeks) | Week 12* | Week 16 (or visit ≥3<br>weeks after week 12) | Response<br>(Confirmed) | Response<br>(unconfirmed) |
|---|---|---|---|---|
| PSA less than baseline | PSA increase that is<br>≥25% and ≥2 ng/mL in<br>absolute value from the<br>nadir (or week 8 visit) | PSA ≥ week 12 visit | PD | PD |
| PSA <u>NOT</u> less<br>than baseline | PSA increase that is<br>≥25% and ≥2 ng/mL in<br>absolute value from the<br>baseline | Any | PD | PD |
| Missing | PSA increase that is ≥25% and ≥2 ng/mL in absolute value from the baseline | PSA ≥ week 12 visit | PD | PD |
| PSA less than baseline | PSA increase that is ≥25% and ≥2 ng/mL in absolute value from the nadir | Results present, PSA < week 12 value (rising trend not confirmed by PSA) | Non-PD | PD |
| PSA less than baseline | PSA increase that is <25% or <2 ng/mL in absolute value from the nadir | Any | Non-PD | Non-PD |
| PSA <u>NOT</u> less<br>than baseline or<br>is missing | PSA increase that is<br><25% or <2 ng/mL in<br>absolute value from the<br>baseline | Any | Non-PD | Non-PD |
| PSA less than baseline | PSA increase that is<br>≥25% and ≥2 ng/mL in<br>absolute value from the<br>nadir (or week 8 visit) | missing | NE | PD |
| Missing | PSA increase that is<br>≥25% and ≥2 ng/mL in<br>absolute value from the<br>baseline | PSA < week 12 visit | Non-PD | PD |
| Missing | PSA increase that is<br>≥25% and ≥2 ng/mL in<br>absolute value from the | missing | NE | PD |

200331

| | Visit | | | |
|---|---|---|---|---|
| Week 8 (or any visit < 12 weeks) | | Week 16 (or visit ≥3<br>weeks after week 12) | | |
| | baseline | | | |
| Results available at week 8 and 12 but do not meet PD definition | | Any | Non-PD | Non-PD |
| If conditions above not met | | Any | NE | NE |

<sup>\* 12</sup> week visit window is defined as follows: If visit occurred under amendment 3, use 78 days  $\pm$  3 days; if visit occurred under amendment 4, use window of 78 days + 5 days.

Note: PSA response of "Any" includes scenarios where results are present and/or missing.

#### 7.2.1.2. Bone Response (at week 12)

The determination of bone response at week 12 is based on PCWG2 criteria for bone progression (Table 2). The algorithm defining the response is outlined in Table 4. The response is categorized into progression (PD), non-PD, not evaluable (NE), and missing.

Table 4 Bone Response Algorithm (based on bone scan results) +

| First post-<br>baseline<br>bone scan<br>prior to 12<br>weeks? | Week 12 visit* | Secondary<br>Assessment (at least<br>6 weeks after week<br>12 visit) | Bone Response<br>(confirmed) | Bone Response<br>(unconfirmed) |
|---|---|---|---|---|
| No | ≥ 2 new lesions | ≥ 2 new lesions | PD | PD |
| No | ≥ 2 new lesions | < 2 new lesions | non-PD | PD |
| No | < 2 new lesions | ≥ 2 new lesions | non-PD | Non-PD |
| No | < 2 new lesions | < 2 new lesions | non-PD | Non-PD |
| No | not done/missing | Any | Not Evaluable | Not Evaluable |
| No | ≥ 2 new lesions | not done/missing | Not Evaluable | PD |
| No | < 2 new lesions | any | Non-PD | Non-PD |
| No | Not done/missing | any | Not Evaluable | Not Evaluable |
| No | not done/missing | not done/missing | Not Evaluable | Not Evaluable |
| Yes | ≥ 2 new lesions | Any (confirmation not required since first bone scan was prior to 12 weeks) | PD | PD |

| First post-<br>baseline<br>bone scan<br>prior to 12<br>weeks? | Week 12 visit* | Secondary<br>Assessment (at least<br>6 weeks after week<br>12 visit) | Bone Response<br>(confirmed) | Bone Response<br>(unconfirmed) |
|---|---|---|---|---|
| Yes | < 2 new lesions | Any | non-PD | Non-PD |
| Yes | not done/missing | Any | Not Evaluable | Not Evaluable |

<sup>\* 12</sup> week visit window is defined as follows: If visit occurred under amendment 3, use 78 days  $\pm$  3 days; if visit occurred under amendment 4, use window of 78 days + 5 days.

#### 7.2.1.3. RECIST Response

The determination of confirmed (and unconfirmed) radiographic response (PR, CR, and PD) at week 12 is based on RECIST v1.1 criteria (Table 1). The algorithm is well defined in the RECIST guidelines (Eisenhauer, 2009). Categories for response include: PD, non-PD (CR, PR, SD, or non-CR/non-PD), NE, and missing (only if no baseline measurable/non-measurable lesions present). The unconfirmed response will also be assessed.

According to PCWG2 criteria, radiological response at week 12 for subjects with baseline disease will be determined by RECIST 1.1 criteria assessed 12 weeks following initiation of GSK2636771 and enzalutamide combination treatment. Since CT/MRI tumour assessments were not scheduled at week 12, the week 16 assessments or the closest unscheduled CT/MRI assessment after week 12 will be used for week 12 RECIST response evaluation.

#### 7.2.1.4. Overall Response (at week 12)

The overall response at week 12 will be used to determine the 12-week non-PD rate. Table 5 provides the algorithm for the derivation of the overall response assessed at 12 weeks post treatment for subjects with or without measurable disease at baseline.

Table 5 Algorithm for Overall Response at Week 12

| Measurable/Non-Measurable<br>Disease Identified at<br>baseline? | RECIST<br>Response<br>(RECIST 1.1) | Bone Response<br>at Week 12 | PSA<br>Response<br>at Week 12 | Overall<br>Response at<br>Week 12<br>(PD/non-<br>PD/NE) |
|---|---|---|---|---|
| Yes | PD | PD | PD | PD |
| Yes | PD | PD | Non-PD | PD |
| Yes | PD | PD | NE | PD |
| Yes | PD | Non-PD | PD | PD |

<sup>\*</sup>This algorithm assumes subjects had bone lesions identified via bone scan at baseline. For subjects without bone lesions identified via Bone Scan at baseline, the confirmed and unconfirmed bone responses are set to missing.

200331

| Measurable/Non-Measurable<br>Disease Identified at<br>baseline? | RECIST<br>Response<br>(RECIST 1.1) | Bone Response<br>at Week 12 | PSA<br>Response<br>at Week 12 | Overall<br>Response at<br>Week 12<br>(PD/non-<br>PD/NE) |
|---|---|---|---|---|
| Yes | PD | Non-PD | Non-PD | PD (via target lesion) |
| Yes | PD | Non-PD | NE | PD (via target lesions) |
| Yes | PD | NE (missing data) | PD | PD |
| Yes | PD | NE (missing data) | Non-PD | PD (via target lesions) |
| Yes | PD | NE (missing data) | NE | PD (via target lesions) |
| Yes | PD | no baseline bone lesions | PD | PD |
| Yes | PD | no baseline bone lesions | Non-PD | PD (via target lesions) |
| Yes | PD | no baseline bone lesions | NE | PD (via target lesions) |
| Yes | Non-PD | PD | PD | PD |
| Yes | Non-PD | PD | Non-PD | PD |
| Yes | Non-PD | PD | NE | PD |
| Yes | Non-PD | Non-PD | PD | Non-PD |
| Yes | Non-PD | Non-PD | Non-PD | Non-PD |
| Yes | Non-PD | Non-PD | NE | Non-PD |
| Yes | Non-PD | NE (missing data) | PD | NE |
| Yes | Non-PD | NE (missing data) | Non-PD | NE |
| Yes | Non-PD | NE (missing data) | NE | NE |
| Yes | Non-PD | no baseline bone lesions | PD | Non-PD |
| Yes | Non-PD | no baseline bone lesions | Non-PD | Non-PD |
| Yes | Non-PD | no baseline bone lesions | NE | Non-PD |
| Yes | NE | PD | PD | PD |
| Yes | NE | PD | Non-PD | PD |
| Yes | NE | PD | NE | PD |
| Yes | NE | Non-PD | PD | NE |
| Yes | NE | Non-PD | Non-PD | NE |
| Yes | NE | Non-PD | NE | NE |
| Yes | NE | NE (missing data) | PD | NE |
| Yes | NE | NE (missing data) | Non-PD | NE |
| Yes | NE | NE (missing data) | NE | NE |
| Yes | NE | no baseline bone | PD | NE |

200331

| Measurable/Non-Measurable Disease Identified at baseline? | RECIST<br>Response<br>(RECIST 1.1) | Bone Response<br>at Week 12 | PSA<br>Response<br>at Week 12 | Overall<br>Response at<br>Week 12<br>(PD/non-<br>PD/NE) |
|---|---|---|---|---|
| | | lesions | | |
| Yes | NE | no baseline bone lesions | Non-PD | NE |
| Yes | NE | no baseline bone lesions | NE | NE |
| No | - | PD | PD | PD |
| No | - | PD | Non-PD | PD |
| No | - | PD | NE | PD |
| No | - | Non-PD | PD | PD |
| No | - | Non-PD | Non-PD | non-PD |
| No | - | Non-PD | NE | non-PD |
| No | - | NE (missing data) | PD | PD |
| No | - | NE (missing data) | Non-PD | Non-PD |
| No | - | NE (missing data) | NE | NE |
| No | - | no baseline bone lesions | PD | PD |
| No | - | no baseline bone lesions | Non-PD | Non-PD |
| No | - | no baseline bone lesions | NE | NE |

Note: "-" = "missing response"

For subjects without measurable/non-measurable disease in baseline, the overall response will be determined on PSA response alone.

Subjects with unknown or missing responses will be treated as having PD (i.e., subjects with NE will be included in the denominator but will not be included in the numerator when calculating the percentage of non-PD).

## 7.2.2. Summary Measure

12 week Non-PD Rate

The number and percentage of participants with the non-PD will be summarized by dose. The corresponding exact 95% Confidence Interval (CI) will also be provided. Subjects with unknown or missing response will be treated as having PD (i.e., subjects with NE will be included in the denominator when calculating the percentage of non-PD).

#### 7.2.3. Population of Interest

The primary efficacy analyses will be based on the All Treated Clinical Activity population, unless otherwise specified. All summaries will be presented by dose, and

overall. The full details of data listings, tables, and figures are presented in Appendix 12: List of Data Displays.

## 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.3. Secondary Efficacy Analyses

## 7.3.1. Endpoint / Variables

PSA and RECIST 1.1 response data will be reported. Subjects with unknown or missing response data, including those who withdraw from the study without an assessment, will be treated as non-responders (i.e., they will be included in the denominator when calculating the percentage). No imputation will be performed for missing lesion assessment or PSA response data. An exact 95% CI will be computed for the PSA50 response rate and RECIST 1.1 confirmed response rate.

Due to the small sample size in the 400 mg cohort (n=2), the radiographic Progression Free Survival (rPFS), time to PSA progression, and time to radiological progression for this cohort will not be summarized separately, however, it will be included in the overall summary. The cohort will also be included in the associated listings.

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

| Secondary<br>Efficacy<br>Endpoint | Definition | Analysis / Display |
|---|---|---|
| PSA50<br>Response<br>Rate | defined as proportion of subjects with a decrease of ≥50% in the PSA concentration from the baseline PSA value determined at least 12 weeks after start of treatment until last post-treatment follow-up visit or initiation of new anti-cancer therapy and confirmed after 3 or more weeks by an additional PSA evaluation. | <ul> <li>Confirmed and unconfirmed PSA changes will be categorized as follows: decline &gt;=50%, PSA increase &gt;=25% (PSA progression per PCWG2), No significant PSA change, and Not Evaluable.</li> <li>Confirmed and unconfirmed PSA50 response rate will be reported by dose level along with the exact 95% confidence interval.</li> <li>See Section 13.6.3 for algorithm details.</li> <li>Waterfall plots will be presented that show the maximum percentage of change in PSA from baseline.</li> <li>Spider plots will be presented to show percent change in PSA from baseline over time</li> </ul> |
| Best Overall<br>Response | defined as the best confirmed/unconfirmed response | Confirmed and unconfirmed best overall response will be reported |

200331

| Secondary<br>Efficacy<br>Endpoint | Definition | Analysis / Display |
|---|---|---|
| (BOR) | (Complete Response [CR] > Partial Response [PR] > Stable Disease [SD] [or non-CR/non-PD] > Progressive Disease [PD] > Not Evaluable [NE]) from combination treatment start date until disease progression or initiation of new anti-cancer therapy, whichever is earlier, as assessed by the investigator per RECIST 1.1 Criteria. | <ul> <li>To be assigned a status of SD, follow-up disease assessment must have met the SD criteria at least once after first dose at a minimum interval of 56 days</li> <li>RECIST 1.1 criteria requires that progression at first assessment be confirmed by a second scan 6 or more weeks later</li> </ul> |
| Objective<br>Response<br>Rate (ORR) | defined as the percentage of subjects with a confirmed complete response (CR) or a partial response (PR) as the BOR, as assessed by the investigator per RECIST 1.1 criteria. | <ul> <li>The number and types of responses, as outlined in RECIST 1.1, will be listed and summarized separately, as appropriate. The investigator observed ORR, confirmed and unconfirmed, will be reported at the interim and final analysis for each cohort specified in treated dose, if data warrant. The estimates along with 95% exact confidence interval (CI) will be provided.</li> <li>Subjects with unknown or missing response will be treated as non-responders, i.e. these subjects will be included in the denominator when calculating the percentage.</li> </ul> |
| | defined as the interval of time (in | The date of disease progression will be defined as the earliest date of disease progression as assessed by the investigator using RECIST 1.1 criteria or progression on bone scan. RECIST 1.1 criteria requires that progression |
| Radiographic<br>Progression-<br>free survival<br>(rPFS) | weeks) between the date of first dose of GSK2636771 and the earlier of the date of disease progression as assessed by the investigator per RECIST 1.1 criteria and the date of death due to any cause. Determination of dates of PFS events and dates for censoring are described in Table 6 | at first assessment be confirmed by a second scan 6 or more weeks later. If no scans are available after the first assessment, the subject should be censored on the date of their first assessment. |
| | | <ul> <li>See Table 1, Bone Response, for definition of<br/>progression on bone scan. Bone progression<br/>at first assessment requires confirmation by a<br/>second scan 6 or more weeks later that<br/>shows a minimum of 2 or more additional new<br/>lesions. If no second scan is available, the<br/>subject should be censored on the date of<br/>their first assessment.</li> </ul> |
| | | rPFS will be summarized by dose level using<br>Kaplan-Meier quantile estimates along with 2-<br>sided 95% CIs. |
| Time to PSA | defined as the time from combination study treatment start | See Table 1 for definition of PSA progression per |

200331

| Secondary<br>Efficacy<br>Endpoint | Definition | Analysis / Display |
|---|---|---|
| progression | until the first PSA progression<br>(confirmed if there has been a<br>PSA decline from baseline) | PCWG2. |
| | | Time to PSA progression will be summarised using Kaplan-Meier methods (plots and summarize table on medians and quartiles) by dose level. |
| Time to radiological progression | | The date of disease progression will be defined as<br>the earliest date of disease progression as<br>assessed by the investigator using RECIST 1.1<br>criteria or progression on bone scan. |
| | defined as the time from | <ul> <li>RECIST 1.1 criteria requires that progression<br/>at first assessment be confirmed by a second<br/>scan 6 or more weeks later. If no scans are<br/>available after the first assessment, the<br/>subject should be censored on the date of<br/>their first assessment.</li> </ul> |
| combination study treatment start until the first radiological progression by RECIST 1.1 and/ or confirmed bone progression. | See Table 1, Bone Response, for definition of progression on bone scan. Bone progression at first assessment by bone scan requires confirmation by a second bone scan 6 or more weeks later that shows a minimum of 2 or more additional new lesions. If no second scan is available, the subject should be censored on the date of their first assessment. | |
| | Time to radiological progression will be<br>summarised using Kaplan-Meier methods (plots<br>and summary table on medians and quartiles) by<br>dose level. | |

200331

## Table 6 Censoring Rules for rPFS Analysis

| Censoring Rules | | |
|---|---|---|
| Scenario | Date of Event (Progression/Death) or Censoring | Event<br>(Progression/Death)<br>or Censoring |
| No adequate baseline tumour assessments (MRI/CT or Bone Scan) and the subject has not died | First Dose Date | Censored |
| No post-baseline tumour assessments and the subject has not died (if the subject has died follow the rules for death indicted at the bottom of the table) | First Dose Date | Censored |
| Progression documented between scheduled visits | Date of assessment of progression <sup>1</sup> | Event |
| With adequate post-baseline assessment and no progression (or death) | Date of last 'adequate' assessment of response <sup>2</sup> | Censored |
| No adequate post-baseline assessment before start of new anticancer therapy | First dose date | censored |
| With adequate post-baseline assessment and new anticancer treatment started (prior to documented disease progression). | Date of last 'adequate' assessment of response <sup>2</sup> (on or prior to starting anticancer therapy) | Censored |
| Death before first PD assessment (or Death at baseline or prior to any adequate assessments) | Date of death | Event |
| Death between adequate assessment visits | Date of death | Event |
| Death or progression after more than one missed visit | Date of last 'adequate' assessment of response <sup>2</sup> (prior to missed assessments)): Since the disease assessment is every 8 weeks, a window of 119 days (16 weeks + 3-day window) will be used to determine whether there is extended time without adequate assessment. If the time difference between PD/death and last adequate disease assessment is more than 119 days, PFS will be censored at the last adequate disease assessment prior to PD/death. | Censored |

#### NOTES:

<sup>&</sup>lt;sup>1</sup> The earliest of (i) Date of radiological assessment showing new lesion (if progression is based on new lesion); or (ii) Date of radiological assessment showing unequivocal progression in non-target lesions, or (iii) Date of last radiological assessment of measured lesions (if progression is based on increase in sum of measured lesions)

<sup>&</sup>lt;sup>2</sup> An adequate assessment is defined as an assessment where the response is CR, PR, or SD.

<sup>&</sup>lt;sup>3</sup> If PD and New anti-cancer therapy occur on the same day, assume the progression was documented first (e.g. outcome is progression and the date is the date of the assessment of progression). If anti-cancer therapy is started prior to any adequate assessments, censoring date should be the date of randomization.

#### 7.3.2. Summary Measure

PSA50 Response Rate

The proportion of subjects with a decrease of  $\geq 50\%$  in the PSA concentration from the baseline PSA value will be categorized as follows: decline  $\geq 50\%$ , PSA increase  $\geq 25\%$  (PSA progression per PCWG2), No significant PSA change, and Not Evaluable. Confirmed and unconfirmed PSA50 response rate will be reported by dose level and overall along with the exact 95% confidence interval. See Section 13.6.3 for algorithm details.

ORR

The number and percentage of participants with the BOR in the following response categories at [timepoint] will be summarized by dose and overall: CR, PR, overall response (CR+PR), SD or Non-CR/Non-PD, PD and NE. The corresponding exact 95% CI for ORR will also be provided. Participants with unknown or missing responses will be treated as non-responders, i.e., these participants will be included in the denominator when calculating percentages of response.

Time to PSA Progression

Time to progression will be summarized descriptively by dose (200 mg and 300 mg doses only) and overall using median(s) and quartiles in the subset of subjects with PSA progression.

Time to Radiological Progression

Time to progression at will be summarized descriptively by dose (200 mg and 300 mg doses only) and overall using median(s) and quartiles in the subset of subjects with radiological progression.

Radiological Progression Free Survival (rPFS)

The distribution of PFS for each dose (200 mg and 300 mg doses only) and overall will be estimated using the Kaplan-Meier method. The median, 25<sup>th</sup> and 75<sup>th</sup> percentiles of PFS will be estimated and corresponding 95% confidence intervals will be estimated using the Brookmeyer-Crowley method (1982). PFS rate and corresponding 95% CI will also be estimated from the Kaplan-Meier analysis.

#### 7.3.3. Population of Interest

The secondary efficacy analyses will be based on the All Treated Clinical Activity population, unless otherwise specified.

#### 7.3.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

200331

Unless otherwise specified, endpoints / variables defined in Section 7.3.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed. No additional statistical analysis will be performed.

#### 8. SAFETY ANALYSES

## 8.1. Overview of Planned Analyses

The safety analyses will be based on the All Treated Safety population, unless otherwise specified, and all summaries and data listings will use treatment labels as specified in Section 5.1. All summaries will be presented by Enzalutamide run-in, combination treatment by dose level, and combination total.

Details of data displays are presented in Appendix 12: List of Data Displays

## 8.2. Extent of Exposure

Dose intensity: Average daily dose on study, cumulative dose of the combination treatment will be summarised with mean, median, standard deviation, minimum, and maximum. The cumulative duration of exposure to the combination treatment in weeks (from first day to last day of treatment plus 1 day) will also be summarised.

Reductions, escalations, and interruptions will be summarised by number of modifications and reasons for modifications for Enzalutamide and GSK2636771 separately. The summaries of dose modifications will be provided only if the data warrant. All the dose reductions, dose escalations and dose interruptions will be listed separately.

## 8.3. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. Details on treatment emergent AEs are provided in Section 13.4.2. Dose modifications (, dose interruptions, dose reductions and dose escalations) and Dose limiting toxicity (DLT) will also be summarized and listed according to GSK Oncology Data Standards.

In addition, a trellis display of subject profiles will be produced that displays individual subject data for renal function tests (correct calcium, magnesium, phosphorous, creatinine, PTH) over time within the same panel for all subjects, along with information regarding age, bone metastasis at baseline, denosumab received within 6 months prior to study, denosumab received during study.

The full details of the planned displays are provided in Appendix 12: List of Data Displays.

## 8.4. Adverse Events of Special Interest (AESI) Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. The list is below:

- Hypocalcaemia
- Increase in Creatinine

## 8.5. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

## 8.6. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. LVEF and Performance status will be summarized and listed based on GSK Oncology Data Standard. The details of the planned displays are presented in Appendix 12: List of Data Displays.

#### 8.6.1. Deaths and Serious Adverse Events

All deaths will be summarised based on the number and percentage of subjects. This summary will classify subjects by time of death relative to the last dose of medication (>30 days or ≤30 days) and primary cause of death (disease under study, SAE related to study treatment, or other). A supportive listing will be generated to provide subject-specific details on subjects who died.

All SAEs will be tabulated based on the number and percentage of subjects who experienced the event. The summary table will be displayed in descending order of total incidence by Preferred Term only.

SAEs will also be summarized by maximum toxicity grade. Relevant serious adverse events will be displayed by preferred term and will be sorted in descending order based on total incidence in each treatment group.

SAEs are included in the listing of all adverse events. Separate supportive listings with subject-level details will be generated for

- Fatal SAEs
- Non-Fatal SAEs.

## 8.7. Pregnancies

A listing of pregnancies will be generated if there was any female partner of the male subjects become pregnant during the study.

#### 9. PHARMACOKINETIC ANALYSES

Pharmacokinetic analysis will be the combined responsibility of GSK Clinical Pharmacology Modelling and Simulation Department and GSK Discovery Biometrics and Clinical Statistics.

The merge of PK concentration data, randomisation and eCRF data will be performed by Clinical Statistics (Programmer).

## 9.1. Primary Pharmacokinetic Analyses

There were no primary pharmacokinetic endpoints defined in the objectives for this study.

## 9.2. Secondary Pharmacokinetic Analyses

#### 9.2.1. Endpoint / Variables

#### 9.2.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.3 Reporting Standards for Pharmacokinetic).

Concentration-time data for GSK2636771, enzalutamide and N-desmethyl enzalutamide from the Dose Escalation Phase will be listed and summarized. In addition, concentration-time figures will be presented.

The following secondary objectives will be displayed graphically:

- The PK of enzalutamide and N-desmethyl enzalutamide following repeat-dose oral administration with and without GSK2636771, and
- The PK of GSK2636771 in the presence of enzalutamide.

#### 9.2.2. Population of Interest

The pharmacokinetic (PK) analyses will be based on the PK Concentration population, unless otherwise specified.

## 9.2.3. Statistical Analyses / Methods

No formal statistical analysis will be performed.
200331

#### 10. BIOMARKER ANALYSES

#### 10.1. Exploratory Biomarker Analyses

#### 10.1.1. Endpoint / Variables

#### 10.1.1.1. Circulating Tumour Cells

CTC response rate will be performed, which is defined as percent of subjects having favourable (CTC <5/7.5 mL of blood) at nadir, if baseline is unfavourable (CTC≥5/7.5mL of blood). Conversions from baseline number of CTCs using the CellSearch platform in blood samples will be summarized and listed as part of this RAP.

If data warrant, additional analysis of CTC will be discussed as part of a RAP supplement; i) Analysis of baseline CTC with clinical outcome (time on treatment and PSA changes

#### 10.1.1.2. Frequency of PTEN loss and Mechanism of PTEN Loss

The frequency of PTEN loss is defined as the proportion of subjects that were tested by central PTEN testing that were identified as PTEN-deficient. The number of tumour biopsy samples with a Histo-score (H score) of 30 and less will be compared with the total number of tumour biopsy samples that were analysed by central PTEN testing to evaluate the frequency of PTEN loss in mCRPC for this study.

The H-Score of all enrolled subjects will be compared to molecular sequencing of tumour biopsy sample to understand the mechanism(/s) of PTEN loss.

#### 10.1.1.3. Mutational Analysis of Tumour Biopsy Sample

Mutational analysis of screening tumour biopsy samples will be analysed to understand gene mutations of mCRPC subjects enrolled in this study and to evaluate the frequency of PTEN homozygous loss. Gene mutations include, small nuclear variant (SNV), copy number variation (gene deletion and gene amplification) and gene fusions.

#### 10.1.2. Summary Measure

- 1. CTC response rate is defined as any conversion from ≥5 at baseline to <5 over the course of the study. Data will be presented as a single line in a table, for each subject.
- 2. PTEN:
  - a. Frequency of PTEN loss by PTEN IHC (H-Score  $\leq$  30) in all screened subjects.
  - b. Homozygous or heterozygous PTEN loss based on Foundation Medicine analysis
- 3. Heatmap representation of all SNV, CNV, gene fusion and indels of genes in the 475 gene panel from Foundation Medicine (n=16 subjects).

200331

## 10.1.3. Population of Interest

The exploratory biomarker analyses will be based on the All Screened and/or Biomarker population, unless otherwise specified.

## 10.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

200331

# 11. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

For this study no on treatment biopsy samples were obtained for Pharmacodynamic analysis. Therefore, no PD analysis can be done for this study.

If data warrant, the pharmacokinetic / pharmacodynamic relationship of GSK2636771 administered in Male Subjects with Metastatic Castration-Resistant Prostate Cancer (mCRPC) may be explored. The influence of subject demographics and baseline characteristics, including disease activity in this population will be investigated.

Further details of PK/PD analyses will be described under a separate RAP. Results of the PK/PD analyses may be included in a report separate from the clinical study report (CSR).

200331

#### 12. REFERENCES

Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics, 1982; 38:29-41.

Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: Revised RECIST guidelines (version 1.1). *European Journal of Cancer*. 2009;45:228-247.

Lee JJ, Liu DD. A predictive probability design for phase II cancer clinical trials. *Clinical Trials*. **5(2)**:93-106. 2008

Scher HI, Halabi S, Tannock I, et al. Design and End Points of Clinical Trials for Patients With Progressive Prostate Cancer and Castrate Levels of Testosterone: Recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008;26:1148-1159.

200331

## 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 13.1.1. Exclusions from Per Protocol Population

No exclusions are noted.

200331

- 13.2. Appendix 2: Schedule of Activities
- 13.2.1. Protocol Defined Schedule of Events
- Table 7 Time and Events Table for Dose Escalation Phase

See following page.

| Study Assessments <sup>1,2</sup> | Pre-Screening | Screening | Enzalutamide<br>Run-In<br>Period | (L | ination Tr | ting Perio | d) | | tment Continuation<br>Period | Time of Discontinuation of Treatment due to Disease Progression31 | Post-Treatment Follow-Up<br>Visit <sup>28</sup> | Extended<br>Follow-Up<br>Visits <sup>29</sup> | Post-<br>Extende<br>d Follow-<br>Up<br>/EOS<br>Visit <sup>30</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day -14<br>to<br>Day -1 | Day 1 to Day<br>14 | Wk 1,<br>Day 1 | Wk 2,<br>Day 8 | Wk 3,<br>Day<br>15 | Wk 4,<br>Day<br>22 | Week<br>5, Day<br>29 | Week 8 and every 4 weeks thereafter | | | Every 3 months | |
| Visit Window | | • | | +1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | +5days Week 12 only;<br>±3 days for all other<br>visits | +1<br>day | -2/+7<br>days | ±14<br>days | ±3<br>days |
| Clinical Assessments | | | | | | | | | | | | | |
| Informed Consent | <b>X</b> 3 | X <sup>4</sup> | | | | | | | | | | | |
| Demographics | Χ | | | | | | | | | | | | |
| Medical History | | Χ | | | | | | | | | | | |
| Determination of PTEN Deficiency Status | M <sup>5</sup> | | | | | | | | | | | | |
| Safety Assessments | | | | | | | | | | | | | |
| ECOG PS | | Х | | Х | | Х | Х | Х | Week 8 and then<br>Q8wks | Х | Χ | | Х |
| Physical Exam | | Х | | Х | | | | | Week 8 and then<br>Q8wks | | Х | | Х |
| Height <sup>8</sup> | | Χ | | | | | | | | | | | |
| Weight | | Х | | Х | | | | | Week 8 and then<br>Q8wks | | Χ | | Х |
| Vital Signs <sup>9</sup> | | Χ | | Χ | Χ | Χ | Χ | Χ | Х | | Χ | | Χ |
| 12-Lead ECG <sup>10</sup> | | X <sub>6</sub> | | Q8wks | | | | Week 8 and then<br>Q8wks | | Х | | Х | |
| ECHO/MUGA | | X6,7 | | As clinically indicated | | | | | | | | | |
| AE Monitoring | | | | Continuous | | | | | X <sup>11</sup> | X <sup>11</sup> | | | |
| Concomitant Medications | | Χ | Continuous | | | | | | | Χ | | | |

| Study Assessments <sup>1,2</sup> | Pre-Screening | Screening | Enzalutamide<br>Run-In<br>Period | (L | ination Ti<br>DLT Repor | rting Perio | d) | | tment Continuation<br>Period | Time of Discontinuation of Treatment due to Disease Progression <sup>31</sup> | Post-Treatment Follow-Up<br>Visit <sup>28</sup> | Extended<br>Follow-Up<br>Visits <sup>29</sup> | Post-<br>Extende<br>d Follow-<br>Up<br>/EOS<br>Visit <sup>30</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day -14<br>to<br>Day -1 | Day 1 to Day<br>14 | Wk 1,<br>Day 1 | Wk 2,<br>Day 8 | Wk 3,<br>Day<br>15 | Wk 4,<br>Day<br>22 | Week<br>5, Day<br>29 | Week 8 and every 4 weeks thereafter | | | Every 3<br>months | |
| Visit Window | | , | | +1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | +5days Week 12 only;<br>±3 days for all other<br>visits | +1<br>day | -2/+7<br>days | ±14<br>days | ±3<br>days |
| Laboratory Assessments | 12 | | | | | | | | | | | | |
| Hematology/<br>Clinical Chemistry | | <b>X</b> 6 | | Χ | Х | Χ | Х | Х | X | | Χ | | Х |
| Ionized Calcium | | <b>X</b> 6 | | X33 | Х | Х | Х | Χ | Х | | Χ | | Χ |
| Vitamin D <sup>34</sup> | | X <sup>6</sup> | | | | | Х | | | | Χ | | Χ |
| Coagulation:<br>PT, PTT, INR | | X <sub>6</sub> | | Х | | | Х | | | | | | |
| Liver function Tests | | <b>X</b> 6 | | Х | Х | Х | Х | Χ | Х | | Χ | | Χ |
| Urinalysis <sup>13</sup> Urine Microscopy <sup>13</sup> UPC <sup>14</sup> | | <b>X</b> 6 | | Х | | | Х | | Х | | Х | | Х |
| Urine Electrolytes <sup>15</sup> | | X <sub>6</sub> | | X33 | | Х | Х | | Week 8 and then<br>Q8wks | | Χ | | |
| Parathyroid Hormone | | | | Χ | | | As clinic | ally indica | ted <sup>16</sup> | | | | |
| Bone Markers <sup>35</sup> | | | | Χ | | | | Х | Weeks 12 and 24 | | Χ | | Χ |
| PSA and LDH32 | | X <sup>6</sup> | | Х | | | | | Х | Х | Χ | | Х |
| Serum Testosterone | | X <sup>6</sup> | | | | | | | | | Χ | | Х |
| PK Assessments | | | | | | | | | | | | | |
| PK Blood Sampling <sup>17</sup> | | | | | | | | Χ | Weeks 8 and 12 | | | | |

| Study Assessments <sup>1,2</sup> | Pre-Screening | Screening | Enzalutamide<br>Run-In<br>Period | (L | ination Ti<br>DLT Repoi | rting Perio | d) | | tment Continuation<br>Period | Time of Discontinuation of Treatment due to Disease Progression31 | Post-Treatment Follow-Up<br>Visit <sup>28</sup> | Extended<br>Follow-Up<br>Visits <sup>29</sup> | Post-<br>Extende<br>d Follow-<br>Up<br>/EOS<br>Visit <sup>30</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day -14<br>to<br>Day -1 | Day 1 to Day<br>14 | Wk 1,<br>Day 1 | Wk 2,<br>Day 8 | Wk 3,<br>Day<br>15 | Wk 4,<br>Day<br>22 | Week<br>5, Day<br>29 | Week 8 and every 4 weeks thereafter | | | Every 3 months | |
| Visit Window | | | | +1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | +5days Week 12 only;<br>±3 days for all other<br>visits | +1<br>day | -2/+7<br>days | ±14<br>days | ±3<br>days |
| Disease Assessments <sup>18</sup> | | | | | | | | | | | | | |
| CT scan or MRI <sup>19</sup> | | X <sup>6,7</sup> | | | | | | | Week 8 and then<br>Q8wks to Week 48;<br>then Q12wks | X | | X | |
| Chest X-ray or Chest CT scan | | X6,7 | | | | | | | | | | | |
| Bone Scan <sup>20</sup> | | X <sup>6,7</sup> | | | | | | | Week 12 and then<br>Q12wks | Х | | Х | |
| Biomarker Assessments | | | | | | | | | | | | | |
| CTC – Janssen <sup>21</sup> | | Χ | | Х | | | Х | | Weeks 8, 16, 24, and 32 | Х | | | |
| CTC – EPIC <sup>22</sup> | | Χ | | | | | | | Week 8 only | Χ | | | |
| Predictive Biomarker:<br>Tumor Tissue <sup>23</sup> | | | | Х | | | | | | | | | |
| Progression Tumor<br>Biopsy <sup>24</sup> | | | | | | | | | | Х | | | |
| Tumor Biopsies for<br>Pharmacodynamics <sup>24</sup> | | | X (Day 14) | | X <sup>24</sup> | | | | | | | | |
| cfDNA/RNA/Soluble<br>Markers <sup>25</sup> | | X | | Х | | | Х | | Weeks 8, 16, 24, and 32 | Х | | | |

200331

| Study Assessments <sup>1,2</sup> | Pre-Screening | Screening | Enzalutamide<br>Run-In<br>Period | | Combination Treatment Period (DLT Reporting Period) | | | Trea | tment Continuation<br>Period | Time of Discontinuation of Treatment due to Disease Progression31 | Post-Treatment Follow-Up<br>Visit <sup>28</sup> | Extended<br>Follow-Up<br>Visits <sup>29</sup> | Post-<br>Extende<br>d Follow-<br>Up<br>/EOS<br>Visit <sup>30</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day -14<br>to<br>Day -1 | Day 1 to Day<br>14 | Wk 1,<br>Day 1 | Wk 2,<br>Day 8 | Wk 3,<br>Day<br>15 | Wk 4,<br>Day<br>22 | Week<br>5, Day<br>29 | Week 8 and every 4 weeks thereafter | | | Every 3 months | |
| Visit Window | | • | | +1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | +5days Week 12 only;<br>±3 days for all other<br>visits | +1<br>day | -2/+7<br>days | ±14<br>days | ±3<br>days |
| Biomarker Assessments | contin | nued | | | | | | | | | | | |
| Blood Sample for<br>Genetic Research <sup>26</sup> | | | | Х | | | | | | | | | |
| Study Treatments <sup>27</sup> | • | | | | | | | | | | | | |
| Enzalutamide | | | Continuous | | • | | Continu | ous | | | • | | |
| GSK2636771 | | | | Continuous | | | ous | | | | | | |

Abbreviations: AE, adverse event; cfDNA, circulating-free tumor DNA; CT, computed tomography; CTC, circulating tumor cells; ECG, electrocardiogram; ECHO, echocardiogram; ECOG, Eastern Cooperative Oncology Group; EOS, End of Study; HbA1C, hemoglobin A1C; INR, international normalization ratio; M, mandatory; MRI, magnetic resonance imaging; MUGA, multigated acquisition scan; O, optional; PD, pharmacodynamics; PK, pharmacokinetics; PS, performance status; PSA, prostate-specific antigen; PT, prothrombin time; PTEN, phosphatase and tensin homolog; PTH, parathyroid hormone; PTT, partial thromboplastin time; Q4wks, every 4 weeks; Q8wks, every 8 weeks; Q12wks, every 12 weeks; UPC, urine:protein:creatinine; Wk(s), week(s)

- 1. **Study Assessments:** All assessments may be performed more frequently if clinically appropriate. Assessments scheduled on days of dosing should be completed prior to the administration of study treatments, unless otherwise specified
- 2. **Study Assessments:** Assessments throughout the study are calendar based starting from Week 1, Day 1 of the Combination Treatment Period (the first dose of combination treatment). Dose interruptions should not alter the assessment schedule for any subsequent treatment period.
- 3. **Pre-Screening Informed Consent:** Separate pre-screening informed consent must be obtained prior to initiation of any pre-screening procedures or assessments.
- 4. Screening Informed Consent: Informed consent must be obtained prior to initiation of any screening procedures or assessments...
- 5. **PTEN Deficiency Status (Mandatory):** Tumor tissue samples (archived or fresh tumor tissue obtained by pre-treatment biopsy) will be collected to determine PTEN deficiency status of the tumor by the designated central laboratory. Refer to the SRM for details about the number of slides to be submitted, preparation, handling and shipping. Results of

- the PTEN deficiency testing from the central laboratory only will be used to determine if the subject is eligible to continue Screening. Only subjects with PTEN deficient tumor based on central laboratory testing results will be screened. Any remaining tumor tissue may be used for other predictive biomarker analyses if consent has been obtained.
- 6. **Screening:** When possible, screening assessments that require imaging, ECG, ECHO/MUGA, or laboratory studies should be performed AFTER PTEN status has been determined.
- 7. **Screening:** All screening assessments must be completed and all entry criteria must be met prior to assessments on Day 1 of Enzalutamide Run-In Period. EXCEPTION: ECHO/MUGA must be completed within 28 days of enrollment (Day 1 of Enzalutamide Run-In Period), and disease assessment must be completed within 28 days (35 days if MRI is used) prior to enrollment (Day 1 of the Enzalutamide Run-In Period).
- 8. **Height** is only measured at Screening.
- 9. Vital Signs: Blood pressure, temperature and heart rate will be measured. Vital signs may be measured more frequently if clinically warranted.
- 10. **ECG:** A single 12-lead ECG is to be performed **before** vital signs are measured and any blood draws, if assessments are planned at the same nominal time point.
- 11. **AE Monitoring:** Continued monitoring of AEs applies only to ongoing events at time of treatment discontinuation.
- 12. **Laboratory Assessments:** Refer to Section 8.6.6 in protocol for list of specific laboratory tests to be performed. Assessments may be performed within 24 hrs prior to scheduled visit (liver function tests and urine tests for UPC may be performed up to 72 hrs prior to a scheduled visit) to ensure availability of results.
- 13. **Urinalysis and Urine Microscopy:** Urinalysis and urine microscopy will be performed at the time points indicated. Assessments may be performed within 24 hrs prior to a scheduled visit to ensure availability of results.
- 14. **UPC:** Urine sample for UPC is to be collected at the time points indicated. Perform UPC with the first morning urine specimen (if possible) when urine dipstick protein ≥2+. Urine samples for UPC may be collected up to 72 hrs prior to a scheduled visit to ensure that results are available at time of visit. If the urine sample collected at Screening is contaminated with other bodily fluids, UPC will not be determined and subject will remain eligible for the study.
- 15. **Urine Electrolytes:** Urine samples will be obtained at Screening, pre-dose on Day 1 (Week 1), Day 3 OR Day 4, Day 15 (Week 3), Day 22 (Week 4) of the Combination Treatment Period, Week 8 and then every 8 weeks (± 3 days) thereafter during the Treatment Continuation Period, and at the post-treatment follow-up visit to determine urine electrolytes (magnesium, phosphorus and calcium) and urine creatinine.
- 16. **Parathyroid Hormone (PTH):** Assessment of PTH will be performed if a Grade 2 or higher hypocalcemia or hypophosphatemia is reported.
- 17. **PK Blood Sampling: Day 14 (Enzalutamide Run-In Period):** Plasma samples for analysis of enzalutamide and N-desmethyl enzalutamide will be collected at pre-dose and 0.5, 1, 2, 3, 4, and 6 hrs post-dose on Day 14 of Enzalutamide Run-In Period, the day prior to administration of the first dose of combination study treatment (GSK2636771 and enzalutamide). **Week 5, Day 29 (Treatment Continuation Period):** Blood and plasma samples for analysis of GSK2636771, enzalutamide and N-desmethyl enzalutamide will be collected at pre-dose and 0.5, 1, 2, 3, 4, and 6 hrs post-dose. Actual date and time of sample collection and dosing of study treatments must be recorded. Explanations are required for any deviations of more than 5 minutes from the planned time during the first 2 hrs and for deviations of more than 20 minutes from the planned time for samples collected at 3 hrs up to 6 hrs post-dose. **Week 8 and Week 12 (Treatment Continuation Period):** Blood and plasma samples for analysis of GSK2636771, enzalutamide and N-desmethyl enzalutamide will be collected pre-dose only.
- 18. **Disease Assessments:** Disease assessments at Screening must be performed within 28 days prior to enrollment (Day 1 of the Enzalutamide Run-In Period), or within 35 days prior to enrollment (Day 1 of the Enzalutamide Run-In Period if disease assessment is performed by MRI, to identify target and non-target lesions.
- 19. **CT scan or MRI:** Scans should be performed at Screening, Week 8 and then every 8 weeks (±7 days) during the first 48 weeks of the Treatment Continuation Period and then every 12 weeks (±7 days) thereafter in the Treatment Continuation Period, and at the time of disease progression. All confirmatory scans are to be performed within 4 weeks (±3 days) of a CR or PR. If a subject discontinues treatment for reasons other than disease progression, disease assessments should continue every 3 months until disease progression, initiation of new anti-cancer treatment, subject withdrawal of consent, or death.
- 20. **Bone Scan:** A bone scan is required for all subjects at Screening. For subjects without bone disease at baseline, subsequent bone scans should be performed as clinically indicated. Subjects with bone metastases at baseline should have a bone scan performed at Week 12 and then every 12 weeks (±7 days) thereafter in the Treatment

- Continuation Period, or as clinically indicated, and at the time of disease progression. If a subject discontinues treatment for reasons other than disease progression, bone scans should continue every 3 months until disease progression, initiation of new anti-cancer treatment, subject withdrawal of consent, or death.
- 21. **CTC-Janssen:** Whole blood samples will be obtained at Screening; pre-dose on Day 1 (Week 1) and Day 22 (Week 4) of the Combination Treatment Period; pre-dose on Day 1 of Weeks 8, 16, 24 and 32 of the Treatment Continuation Period; and at time of disease progression.
- 22. **CTC-EPIC:** Whole blood samples will be obtained at Screening, pre-dose on Day 1 of Week 8 of the Treatment Continuation Period, and at the time of disease progression for protein and genomic analysis.
- 23. **Predictive Biomarkers Tumor Tissue:** For subjects enrolled into the study, additional slides of tumor tissue samples will be collected and submitted to the designated laboratory for analysis once a subject has received their first dose of GSK2636771 on Week 1, Day 1 of the Combination Treatment Period. Tumor tissue may be obtained from archived tissue samples or fresh tumor tissue submitted for the PTEN testing. If additional tumor tissue is not available, no new biopsy procedure is required for predictive biomarker analysis. Refer to the SRM for details about the number of slides to be submitted, preparation, handling and shipping.
- 24. **Tumor Biopsies for PD and progression**: These biopsies are optional and may be undertaken in select cases upon agreement with the investigator and when consent is provided by the subject. For pharmacodynamic biomarker analyses, fresh tissue biopsies would be collected between Day 12 of the Enzalutamide Run-in Period and Week 1/Day 1, prior to any treatment with GSK2636771, and 2-4 hours post dose between Days 8 and 15 of the Combination Treatment Period (post-treatment). For subjects who consent to the optional progression biopsy, a fresh tumor biopsy should be completed if the subject initially responded to combination treatment and then progressed.
- 25. **cfDNA/RNA/Soluble Markers:** Plasma samples will be obtained from collected blood samples at Screening, pre-dose on Weeks 1, 4, 8, 16, 24, and 32 of the Combination Treatment Period, and at the time of treatment discontinuation due to disease progression. Plasma will be analyzed for genomic changes in the circulating tumor DNA, RNA, and soluble markers.
- 26. **Genetic Research:** A 6-mL blood sample should be collected after Screening, preferably on Week 1, Day 1 of the Combination Treatment Period, if informed consent has been obtained for genetic research.
- 27. **Study Treatment:** Enzalutamide monotherapy should be taken once daily during the Enzalutamide Run-In Period. Enzalutamide will be self-administered in the clinic on Day 14 of the Enzalutamide Run-In Period. GSK2636771 and enzalutamide will be administered in the clinic on Week 1, Day 1 of the Combination Treatment Period and on days when blood, plasma, and/or urine samples are collected for analysis of PK, CTC, and/or urine electrolytes.
- 28. **Post-Treatment Follow-Up Visit:** *ONLY* subjects who withdraw during the Enzalutamide Run-In Period or withdraw from study treatment *due to* disease progression (see Section 5.2 in protocol) should have a post-treatment follow-up visit conducted within approximately 30 days (-2/+7 days) of last dose of study treatment(s). If a subject is unable to return to the clinic due to hospitalization, site staff is encouraged to call subject for assessment of AEs.
- 29. **Extended Follow-Up Visits:** Subjects who withdraw from study treatment *without* disease progression should be contacted every 3 months (±14 days) until disease progression, death, withdrawal of consent, or subject is lost to follow-up. Contact may include a clinic visit, a telephone contact, or an e-mail. The initiation of any new anti-cancer treatments and date of last contact should be documented.
- 30. Post-Extended Follow-Up/EOS Visit: ONLY subjects who discontinue the Extended Follow-Up Visits should have a Post-Extended Follow-Up/EOS Visit performed.
- 31. Subjects are not required to discontinue treatment on the basis of PSA progression alone or for the worsening of an isolated disease site that is not clinically significant (see Section 5.2 in protocol)
- 32. When collected as part of the routine standard of care for a subject, LDH will be reported.
- 33. Complete clinical chemistries laboratory assessments at Week1/Day 1 and **again on either Day 3 or Day 4**. The Day 3 or Day 4 assessments can be completed at a local laboratory and does **not** require a clinic visit. The hematology panel does NOT need to be collected on Day 3/ Day.4. Review of these labs must occur before Week 2, Day 1 visit.
- 34. Includes assessments for 25-OH D and 1,25-OH2 D.
- 35. Includes urine and blood and/or serum samples. Must be collected at the same time of day (±1 hour) to eliminate diurnal effects, and after fasting. See SRM for additional details on the specific assessments and sample collection.

200331

## Table 8 Time and Events Table for Dose Expansion Phase

See following page.

| Study Assessments <sup>1,2</sup> | Pre-Screening | Screening | Enzalutamide<br>Run-In<br>Period | (L | Combination Treatment Period (DLT Reporting Period) Treatment Continuation Period | | | Time of Discontinuation of Treatment due to Disease Progression <sup>31</sup> | Post-Treatment Follow-Up<br>Visit <sup>28</sup> | Extended<br>Follow-Up<br>Visits <sup>29</sup> | Post-<br>Extended<br>Follow-Up<br>/EOS<br>Visit <sup>30</sup> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day -14<br>to<br>Day -1 | Day 1 to Day<br>14 | Wk 1,<br>Day 1 | Wk 2,<br>Day 8 | Wk 3,<br>Day<br>15 | Wk 4,<br>Day<br>22 | Week<br>5, Day<br>29 | Week 8 and every 4 weeks thereafter | | | Every 3<br>months | |
| Visit Window | | | | +1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | +5days Week 12 only;<br>±3 days for all other<br>visits | +1<br>day | -2/+7<br>days | ±14<br>days | ±3<br>days |
| Clinical Assessments | | | | | | | | | | | | | |
| Informed Consent | <b>X</b> 3 | X <sup>4</sup> | | | | | | | | | | | |
| Demographics | Χ | | | | | | | | | | | | |
| Medical History | | Χ | | | | | | | | | | | |
| Determination of PTEN Deficiency Status | M <sup>5</sup> | | | | | | | | | | | | |
| Safety Assessments | | | | | | | | | | | | | |
| ECOG PS | | Х | | Х | | Х | Х | Х | Week 8 and then<br>Q8wks | Х | Х | | Х |
| Physical Exam | | Х | | Х | | | | | Week 8 and then<br>Q8wks | | Х | | Х |
| Height <sup>8</sup> | | Χ | | | | | | | | | | | |
| Weight | | Х | | Х | | | | | Week 8 and then<br>Q8wks | | Х | | Х |
| Vital Signs <sup>9</sup> | | Χ | | Χ | Х | Х | Χ | Χ | Х | | Χ | | Х |
| 12-Lead ECG <sup>10</sup> | | X <sub>6</sub> | | | | | Χ | | Week 8 and then<br>Q8wks | | Χ | | X |
| ECHO/MUGA | | X6,7 | | As clinically indicated | | | | | | | | | |
| AE Monitoring | | | | Continuous | | | | | | X <sup>11</sup> | X <sup>11</sup> | | |
| Concomitant Medications | | Χ | | Continuous | | | | | | | Χ | | |

| Study Assessments <sup>1,2</sup> | Pre-Screening | Screening | Enzalutamide<br>Run-In<br>Period | (L | OLT Repo | reatment<br>rting Perio | d) | | tment Continuation<br>Period | Time of Discontinuation of<br>Treatment due to Disease<br>Progression <sup>31</sup> | Post-Treatment Follow-Up<br>Visit <sup>28</sup> | Extended<br>Follow-Up<br>Visits <sup>29</sup> | Post-<br>Extended<br>Follow-Up<br>/EOS<br>Visit <sup>30</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day -14<br>to<br>Day -1 | Day 1 to Day<br>14 | Wk 1,<br>Day 1 | Wk 2,<br>Day 8 | Wk 3,<br>Day<br>15 | Wk 4,<br>Day<br>22 | Week<br>5, Day<br>29 | Week 8 and every 4 weeks thereafter | | | Every 3<br>months | |
| Visit Window | | , | | +1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | +5days Week 12 only;<br>±3 days for all other<br>visits | +1<br>day | -2/+7<br>days | ±14<br>days | ±3<br>days |
| Laboratory Assessments | 12 | | | | | | | | | | | | |
| Haematology/ Clinical Chemistry | | <b>X</b> 6 | | Х | Х | X | Х | Х | X | | Х | | Х |
| Ionized Calcium | | X <sup>6</sup> | | X33 | Х | Х | Х | Х | Х | | Χ | | Х |
| Vitamin D <sup>34</sup> | | X6 | | | | | Х | | | | Х | | Х |
| Coagulation:<br>PT, PTT, INR | | X <sup>6</sup> | | Х | | | Х | | | | | | |
| Liver function Tests | | <b>X</b> 6 | | Χ | Χ | Х | Χ | Х | X | | Χ | | X |
| Urinalysis <sup>13</sup> Urine Microscopy <sup>13</sup> UPC <sup>14</sup> | | X6 | | Х | | | Х | | Х | | Х | | Х |
| Urine Electrolytes <sup>15</sup> | | X6 | | X33 | | Х | Х | | Week 8 and then<br>Q8wks | | Х | | |
| Parathyroid Hormone | | | | Х | | | As clinic | ally indica | | | | | |
| Bone Markers <sup>35</sup> | | | | Χ | | | | Х | Weeks 12 and 24 | | Χ | | Х |
| PSA and LDH <sup>32</sup> | | X <sup>6</sup> | | Χ | | | | | X | Х | Χ | | X |
| Serum Testosterone | | X <sub>6</sub> | | | | | | | | | Χ | | Х |
| PK Assessments | | | ı | | | | 1 | | | | | 1 | |
| PK Blood Sampling <sup>17</sup> | | | | | | | | X | Weeks 8 and 12 | | | | |

| Study Assessments <sup>1,2</sup> | Pre-Screening | Screening | Enzalutamide<br>Run-In<br>Period | (L | OLT Repo | r <b>eatment</b><br>rting Perio | d) | | tment Continuation<br>Period | Time of Discontinuation of Treatment due to Disease Progression <sup>31</sup> | Post-Treatment Follow-Up<br>Visit <sup>28</sup> | Extended<br>Follow-Up<br>Visits <sup>29</sup> | Post-<br>Extended<br>Follow-Up<br>/EOS<br>Visit <sup>30</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day -14<br>to<br>Day -1 | Day 1 to Day<br>14 | Wk 1,<br>Day 1 | Wk 2,<br>Day 8 | Wk 3,<br>Day<br>15 | Wk 4,<br>Day<br>22 | Week<br>5, Day<br>29 | Week 8 and every 4 weeks thereafter | | | Every 3<br>months | |
| Visit Window | | • | | +1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | +5days Week 12 only;<br>±3 days for all other<br>visits | +1<br>day | -2/+7<br>days | ±14<br>days | ±3<br>days |
| Disease Assessments <sup>18</sup> | | | | | | | | | | | | | |
| CT scan or MRI <sup>19</sup> | | X <sup>6,7</sup> | | | | | | | Week 8 and then<br>Q8wks to Week 48;<br>then Q12wks | Х | | X | |
| Chest X-ray or Chest CT scan | | X6,7 | | | | | | | | | | | |
| Bone Scan <sup>20</sup> | | X6,7 | | | | | | | Week 12 and then<br>Q12wks | Х | | Х | |
| Biomarker Assessments | | | | | | | | | | | | | |
| CTC – Janssen <sup>21</sup> | | Х | | Х | | | Х | | Weeks 8, 16, 24, and 32 | Х | | | |
| CTC – EPIC <sup>22</sup> | | Χ | | | | | | | Week 8 only | Х | | | |
| Predictive Biomarker:<br>Tumor Tissue <sup>23</sup> | | | | Х | | | | | | | | | |
| Progression Tumor<br>Biopsy <sup>24</sup> | | | | | | | | | | Х | | | |
| Tumor Biopsies for Pharmacodynamics <sup>24</sup> | | | X (Day 14) | | X <sup>24</sup> | | | | | | | | |
| cfDNA/RNA/Soluble<br>Markers <sup>25</sup> | | Х | | Х | | | Х | | Weeks 8, 16, 24, and 32 | Х | | | |

200331

| Study Assessments <sup>1,2</sup> | Pre-Screening | Screening | Enzalutamide<br>Run-In<br>Period | (L | Combination Treatment Period (DLT Reporting Period) Treatment Continuation Period | | Time of Discontinuation of<br>Treatment due to Disease<br>Progression <sup>31</sup> | Post-Treatment Follow-Up<br>Visit <sup>28</sup> | Extended<br>Follow-Up<br>Visits <sup>29</sup> | Post-<br>Extended<br>Follow-Up<br>/EOS<br>Visit <sup>30</sup> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day -14 | Day 1 to Day | Wk 1, | Wk 2, | Wk 3, | Wk 4, | Week | Week 8 and every 4 | | | Every 3 | |
| | | to | 14 | Day 1 | Day 8 | Day | Day | 5, Day | weeks thereafter | | | months | |
| | | Day -1 | | | | 15 | 22 | 29 | | | | | |
| Visit Window | | | | +1 | <u>±</u> 1 | <u>±</u> 1 | <u>±</u> 1 | <u>±</u> 1 | +5days Week 12 only; | +1 | -2/+7 | <u>+</u> 14 | <u>+</u> 3 |
| | | | | day | day | day | day | day | $\pm 3$ days for all other | day | days | days | days |
| | | | | | | | | | visits | | | | |
| Biomarker Assessments | contin | nued | | | | | | | | | | | |
| Blood Sample for | | | | Χ | | | | | | | | | |
| Genetic Research <sup>26</sup> | | | | | | | | | | | | | |
| Study Treatments <sup>27</sup> | | | | | | | | | | | | | |
| Enzalutamide | | | Continuous | | | | Continu | ous | | | | | |
| GSK2636771 | | | | Continuou | | | ous | | | | | | |

Abbreviations: AE, adverse event; cfDNA, circulating-free tumor DNA; CT, computed tomography; CTC, circulating tumor cells; ECG, electrocardiogram; ECHO, echocardiogram; ECOG, Eastern Cooperative Oncology Group; EOS, End of Study; HbA1C, hemoglobin A1C; INR, international normalization ratio; M, mandatory; MRI, magnetic resonance imaging; MUGA, multigated acquisition scan; O, optional; PD, pharmacodynamics; PK, pharmacokinetics; PS, performance status; PSA, prostate-specific antigen; PT, prothrombin time; PTEN, phosphatase and tensin homolog; PTH, parathyroid hormone; PTT, partial thromboplastin time; Q4wks, every 4 weeks; Q8wks, every 8 weeks; Q12wks, every 12 weeks; UPC, urine:protein:creatinine; Wk(s), week(s)

- 1. **Study Assessments:** All assessments may be performed more frequently if clinically appropriate. Assessments scheduled on days of dosing should be completed prior to the administration of study treatments, unless otherwise specified
- 2. **Study Assessments:** Assessments throughout the study are calendar based starting from Week 1, Day 1 of the Combination Treatment Period (the first dose of combination treatment). Dose interruptions should not alter the assessment schedule for any subsequent treatment period.
- 3. **Pre-Screening Informed Consent:** Separate pre-screening informed consent must be obtained prior to initiation of any pre-screening procedures or assessments.
- 4. Screening Informed Consent: Informed consent must be obtained prior to initiation of any screening procedures or assessments...
- 5. **PTEN Deficiency Status (Mandatory):** Tumor tissue samples (archived or fresh tumor tissue obtained by pre-treatment biopsy) will be collected to determine PTEN deficiency status of the tumor by the designated central laboratory. Refer to the SRM for details about the number of slides to be submitted, preparation, handling and shipping. Results of

- the PTEN deficiency testing from the central laboratory only will be used to determine if the subject is eligible to continue Screening. Only subjects with PTEN deficient tumor based on central laboratory testing results will be screened. Any remaining tumor tissue may be used for other predictive biomarker analyses if consent has been obtained.
- 6. **Screening:** When possible, screening assessments that require imaging, ECG, ECHO/MUGA, or laboratory studies should be performed AFTER PTEN status has been determined.
- 7. **Screening:** All screening assessments must be completed and all entry criteria must be met prior to assessments on Day 1 of Enzalutamide Run-In Period. EXCEPTION: ECHO/MUGA must be completed within 28 days of enrollment (Day 1 of Enzalutamide Run-In Period), and disease assessment must be completed within 28 days (35 days if MRI is used) prior to enrollment (Day 1 of the Enzalutamide Run-In Period).
- 8. **Height** is only measured at Screening.
- 9. Vital Signs: Blood pressure, temperature and heart rate will be measured. Vital signs may be measured more frequently if clinically warranted.
- 10. **ECG:** A single 12-lead ECG is to be performed **before** vital signs are measured and any blood draws, if assessments are planned at the same nominal time point.
- 11. **AE Monitoring:** Continued monitoring of AEs applies only to ongoing events at time of treatment discontinuation.
- 12. **Laboratory Assessments:** Refer to Section 8.6.6 in protocol) for list of specific laboratory tests to be performed. Assessments may be performed within 24 hrs prior to scheduled visit (liver function tests and urine tests for UPC may be performed up to 72 hrs prior to a scheduled visit) to ensure availability of results.
- 13. **Urinalysis and Urine Microscopy:** Urinalysis and urine microscopy will be performed at the time points indicated. Assessments may be performed within 24 hrs prior to a scheduled visit to ensure availability of results.
- 14. **UPC:** Urine sample for UPC is to be collected at the time points indicated. Perform UPC with the first morning urine specimen (if possible) when urine dipstick protein ≥2+. Urine samples for UPC may be collected up to 72 hrs prior to a scheduled visit to ensure that results are available at time of visit. If the urine sample collected at Screening is contaminated with other bodily fluids, UPC will not be determined and subject will remain eligible for the study.
- 15. **Urine Electrolytes:** Urine samples will be obtained at Screening, pre-dose on Day 1 (Week 1), Day 3 OR Day 4, Day 15 (Week 3), Day 22 (Week 4) of the Combination Treatment Period, Week 8 and then every 8 weeks (± 3 days) thereafter during the Treatment Continuation Period, and at the post-treatment follow-up visit to determine urine electrolytes (magnesium, phosphorus and calcium) and urine creatinine.
- 16. **Parathyroid Hormone (PTH):** Assessment of PTH will be performed if a Grade 2 or higher hypocalcemia or hypophosphatemia is reported.
- 17. **PK Blood Sampling: Week 5, Day 29 (Treatment Continuation Period):** Blood and plasma samples for analysis of GSK2636771, enzalutamide and N-desmethyl enzalutamide will be collected at pre-dose and 1, 2, and 3 hrs post-dose if a morning clinic visit is scheduled, or at approximately 5 to 6, 6 to 7, and 7 to 8 hrs post-dose if an afternoon clinic visit is scheduled. Actual date and time of sample collection and dosing of study treatments must be recorded. Explanations are required for any deviations of more than 5 minutes from the planned time during the first 2 hrs and for deviations of more than 20 minutes from the planned time for samples collected at 3 hrs up to 8 hrs post-dose. **Week 8 and Week 12 (Treatment Continuation Period):** Blood and plasma samples for analysis of GSK2636771, enzalutamide and N-desmethyl enzalutamide will be collected predose only.
- 18. **Disease Assessments:** Disease assessments at Screening must be performed within 28 days prior to enrollment (Day 1 of the Enzalutamide Run-In Period), or within 35 days prior to enrollment (Day 1 of the Enzalutamide Run-In Period if disease assessment is performed by MRI, to identify target and non-target lesions.
- 19. **CT scan or MRI:** Scans should be performed at Screening, Week 8 and then every 8 weeks (±7 days) during the first 48 weeks of the Treatment Continuation Period and then every 12 weeks (±7 days) thereafter in the Treatment Continuation Period, and at the time of disease progression. All confirmatory scans are to be performed within 4 weeks (±3 days) of a CR or PR. If a subject discontinues treatment for reasons other than disease progression, disease assessments should continue every 3 months until disease progression, initiation of new anti-cancer treatment, subject withdrawal of consent, or death.
- 20. **Bone Scan:** A bone scan is required for all subjects at Screening. For subjects without bone disease at baseline, subsequent bone scans should be performed as clinically indicated. Subjects with bone metastases at baseline should have a bone scan performed at Week 12 and then every 12 weeks (±7 days) thereafter in the Treatment

- Continuation Period, or as clinically indicated, and at the time of disease progression. If a subject discontinues treatment for reasons other than disease progression, bone scans should continue every 3 months until disease progression, initiation of new anti-cancer treatment, subject withdrawal of consent, or death.
- 21. **CTC-Janssen:** Whole blood samples will be obtained at Screening; pre-dose on Day 1 (Week 1) and Day 22 (Week 4) of the Combination Treatment Period; pre-dose on Day 1 of Weeks 8, 16, 24 and 32 of the Treatment Continuation Period; and at time of disease progression.
- 22. **CTC-EPIC:** Whole blood samples will be obtained at Screening, pre-dose on Day 1 of Week 8 of the Treatment Continuation Period, and at the time of disease progression for protein and genomic analysis.
- 23. **Predictive Biomarkers Tumor Tissue:** For subjects enrolled into the study, additional slides of tumor tissue samples will be collected and submitted to the designated laboratory for analysis once a subject has received their first dose of GSK2636771 on Week 1, Day 1 of the Combination Treatment Period. Tumor tissue may be obtained from archived tissue samples or fresh tumor tissue submitted for the PTEN testing. If additional tumor tissue is not available, no new biopsy procedure is required for predictive biomarker analysis. Refer to the SRM for details about the number of slides to be submitted, preparation, handling and shipping.
- 24. **Tumor Biopsies for PD and progression**: These biopsies are optional and may be undertaken in select cases upon agreement with the investigator and when consent is provided by the subject. For pharmacodynamic biomarker analyses, fresh tissue biopsies would be collected between Day 12 of the Enzalutamide Run-in Period and Week 1/Day 1, prior to any treatment with GSK2636771, and 2-4 hours post dose between Days 8 and 15 of the Combination Treatment Period (post-treatment). For subjects who consent to the optional progression biopsy, a fresh tumor biopsy should be completed if the subject initially responded to combination treatment and then progressed..
- 25. **cfDNA/RNA/Soluble Markers:** Plasma samples will be obtained from collected blood samples at Screening, pre-dose on Weeks 1, 4, 8, 16, 24, and 32 of the Combination Treatment Period, and at the time of discontinuation of treatment due to disease progression. Plasma will be analyzed for genomic changes in the circulating tumor DNA, RNA, and soluble markers.
- 26. **Genetic Research:** A 6-mL blood sample should be collected after Screening, preferably on Week 1, Day 1 of the Combination Treatment Period, if informed consent has been obtained for genetic research.
- 27. **Study Treatment:** Enzalutamide monotherapy should be taken once daily during the Enzalutamide Run-In Period. Enzalutamide will be self-administered in the clinic on Day 14 of the Enzalutamide Run-In Period. GSK2636771 and enzalutamide will be administered in the clinic on Week 1, Day 1 of the Combination Treatment Period and on days when blood, plasma, and/or urine samples are collected for analysis of PK, CTC, and/or urine electrolytes.
- 28. **Post-Treatment Follow-Up Visit:** *ONLY* subjects who withdraw during the Enzalutamide Run-In Period or withdraw from study treatment *due to* disease progression see Section 5.2 in protocol) should have a post-treatment follow-up visit conducted within approximately 30 days (-2/+7 days) of last dose of study treatment(s). If a subject is unable to return to the clinic due to hospitalization, site staff is encouraged to call subject for assessment of AEs.
- 29. **Extended Follow-Up Visits:** Subjects who withdraw from study treatment *without* disease progression should be contacted every 3 months (±14 days) until disease progression, death, withdrawal of consent, or subject is lost to follow-up. Contact may include a clinic visit, a telephone contact, or an e-mail. The initiation of any new anti-cancer treatments and date of last contact should be documented.
- 30. Post-Extended Follow-Up/EOS Visit: ONLY subjects who discontinue the Extended Follow-Up Visits should have a Post-Extended Follow-Up/EOS Visit performed.
- 31. These assessments should be completed at the time of disease progression that leads to discontinuation of treatment. Subjects are not required to discontinue treatment on the basis of PSA progression alone or for the worsening of an isolated disease site that is not clinically significant (see Section 5.2 in protocol).
- 32. When collected as part of the routine standard of care for a subject, LDH will be reported.
- 33. Complete clinical chemistries laboratory assessments at Week1/Day 1 and **again on either Day 3 or Day 4**. The Day 3 or Day 4 assessments can be completed at a local laboratory and does **not** require a clinic visit. The hematology panel does NOT need to be collected on Day 3/ Day.4. Review of these labs must occur before Week 2, Day 1 visit.
- 34. Includes assessments for 25-OH D and 1,25-OH2 D.
- 35. Includes urine and blood and/or serum samples. Must be collected at the same time of day (±1 hour) to eliminate diurnal effects, and after fasting. See SRM for additional details on the specific assessments and sample collection

200331

## 13.3. Appendix 3: Assessment Windows

## 13.3.1. Definitions of Assessment Windows for Analyses

| Analysis Set | Parameter | Target | Analysis | Window | Analysis |
|---|---|---|---|---|---|
| / Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| Primary/Seco<br>ndary Efficacy | For patients<br>seen at week<br>12 under<br>protocol<br>amendment 1-3 | Week 12 $\pm$ 3 days | 78-3 days | 78 + 3 days | Week 12 |
| Primary/Seco<br>ndary Efficacy | For patients<br>seen at week<br>12 under<br>protocol<br>amendment 4 | Week 12 + 5 days | 78 days | 78+5 days | Week 12 |

200331

## 13.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 13.4.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | End Date < Combination Treatment Start Date |
| Post-Treatment | Start Date > Stop Date of GSK2636771 |
| | For interim analyses when subjects are still on treatment, Study Treatment Stop Date will be imputed following rules specified in Section 13.7.2.1. |
| Concomitant | Any medication that is not a prior or post -treatment |

#### NOTES:

• Please refer to Section 13.7.2.1: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

#### 13.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | If AE onset date is on or after treatment start date or missing &: |
| Emergent | <ul> <li>Treatment Start Date≤ AE Start Date AE start data is missing</li> </ul> |

#### NOTES:

- Treatment start date refers to the time the first dose of enzalutamide is administered on Day 1 of the Enzalutamide Run-In Period
- Treatment stop date refers to the date of discontinuation of study treatments(s)
- If the treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

200331

## 13.5. Appendix 5: Data Display Standards & Handling Conventions

#### 13.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | , ,, |
| HARP Server | : US1SALX00259 |
| HARP Compound | : arprod\gsk2636771\mid200331\ |
| Analysis Datasets | |
| Analysis datasets | will be created according to IDSL standard. |
| Generation of RTF Files | |
| RTF files will be generated for all tables | |

#### 13.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
   For worst-case analysis, unscheduled visits will be included.
- All unscheduled visits will be included in listings.

200331

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 13.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to [Insert document name]. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Not applicable. |
| NONMEM/PK/PD<br>File | Not applicable. |

200331

#### 13.6. Appendix 6: Derived and Transformed Data

#### 13.6.1. General

#### Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 13.3.1), the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day for Safety**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Date ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### Study Day for Efficacy

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing

- → Study Day = Missing
- Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
- Ref Date ≥ First Dose Date → Study Day = Ref Date First Dose Date + 1

#### **Change from Baseline**

- Change from Baseline = Post-Baseline Visit Value Baseline
- % Change from Baseline = 100 x (Post-Baseline Visit Value Baseline) / Baseline
- Maximum Increase/Decrease from Baseline = maximum (Increase/Decrease from Baseline)
- If either the Baseline or Post-Baseline Visit Value is missing, Change from Baseline and % Change from Baseline is set to missing

#### **Date of Response**

For post-baseline disease assessments, the date of response (PR or better) is assigned to the latest
date of disease assessments; for other response categories (SD or Non-CR/Non-PD, NE, PD), the date
of response is assigned to the earliest date of disease assessments.

#### **Date of New Anti-Cancer Therapy**

 Derived as the earliest date of new anti-cancer therapy, radiotherapy (where applicable) or cancerrelated surgical procedure (where applicable). Missing or partial dates will be imputed for derivation of new anti-cancer therapy following rules specified in Section 13.7.2.1.

200331

#### 13.6.2. Study Population

#### **Treatment Compliance**

Treatment compliance will be calculated based on the formula:

## Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

- Frequency is 2 for BID and 1 for QD. Treatment compliance could be greater than 100% if there are
  events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.
- Planned Treatment Duration is defined as the time from start of study treatment until treatment end date.

#### **Extent of Exposure**

- Missing treatment stop date will be imputed following rules specified in Section 13.7.2.1.
- Daily Oral Drugs
  - Extent of exposure will be calculated for each treatment component
  - Number of days of exposure (duration on study treatment) to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - Treatment Start Date + 1

- Participants who were assigned a treatment but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### **Time since Initial Diagnosis**

- Calculated as the number of [Days] from the Date of Initial Diagnosis:
  - [Randomization/First Dose Date] = Missing
     → Elapse Time = Missing
  - Date of Initial Diagnosis = Completely/partially Missing → Elapse Time = Missing
  - Otherwise → Elapse Time = [Randomization/First Dose Date] Date of Initial Diagnosis + 1

#### 13.6.3. **Efficacy**

#### PSA response (including PSA50 response)

- Using the following algorithm, the following 4 categories will be created:
  - [PSA] Decline>=50% from baseline [confirmed/unconfirmed] (PSA50)
  - No significant PSA change
  - PSA Progression (PSA increase >=25% from baseline)
  - Not Evaluable
- For at least 12 weeks PSA: for visits under amendment 3, use week  $12 \pm 3$  days; for visits under amendment 4, use week 12 + 5 days

#### PSA Response Algorithm – PSA50 unconfirmed

- Step 1: Within identified population define PSA Analysis Set
  - If there is no post-baseline PSA visit with a non-missing result, output to [Not Evaluable]
  - If there is no baseline PSA, output to [Not Evaluable]
  - Output rest to [PSA evaluable Analysis Set]
- Step 2: within [PSA evaluable Analysis Set] create two subsets
  - If any post-baseline visit PSA < baseline output to subset I (decline from baseline)
  - Else if the visit is post-baseline output to Subset II (no decline from baseline)

200331

#### PSA response (including PSA50 response)

- Step 3. Under Subset I:
  - For each subject retain the response flag (urspflg). Find the first visit PSA <= 0.5\*baseline, add urspflg (unconfirmed PSA response flag) =1; output to [Decline>=50% from baseline (unconfirmed]
  - Else output to [temp set 1]
  - Among [temp set 1], find nadir (lowest PSA value at this or any earlier visit through baseline)
     Retain nadir for each subject.
    - PSA >=1.25\*nadir and (PSA-nadir)>=2ng/mL, add uprgflg (unconfirmed PSA progression flag)=1
    - If PSA >=1.25\*nadir and (PSA-nadir)≥ 2ng/mL is confirmed by a second PSA value obtained >=21 days (3 weeks) from the initial increase, add cprgflg (confirmed PSA progression flag)=1
  - If progression is confirmed [sum(uprgflg,cprgflg)=2] output to [PSA progression]
  - Else output to [No significant PSA change]
- Step 4. Under Subset II
  - If any visit >=XX days (12 weeks) PSA >= 1.25\*baseline and abs(increase from baseline) >=2ng/mL output to [PSA progression] (no confirmation required).
  - Else output to [No significant PSA change]

#### PSA Response Algorithm - PSA50 Confirmed

#### NOTE: Steps are very similar to unconfirmed PSA50 with differences indicated in Red.

- Step 1: Within identified population define PSA Analysis Set
  - If there is no post-baseline PSA visit with a non-missing result, output to [Not Evaluable]
  - If there is no baseline PSA, output to [Not Evaluable]
  - Output rest to [PSA evaluable Analysis Set]
- Step 2: within [PSA evaluable Analysis Set] create two subsets
  - If any post-baseline visit PSA < baseline output to subset I (decline from baseline)
  - Else if the visit is post-baseline output to Subset II (no decline from baseline)
- Step 3. Under Subset I:
  - For each subject retain the response flags (urspflg and crspflg). Find the first visit PSA <= 0.5\*baseline, add urspflg (unconfirmed PSA response flag) =1;</li>
  - Find the second visit PSA <= 0.5\*baseline, if this visit time is >=21 days (3 weeks) from the first visit, add crspflg (confirmed PSA response flag)=1
  - If the response is confirmed (urspflg+crspflg)=2, output to [Decline>=50% from baseline (confirmed)
  - Else output to [temp set 1]
  - Among [temp set 1], find nadir (lowest PSA value at this or any earlier visit through baseline)
     Retain nadir for each subject.
    - PSA >=1.25\*nadir and (PSA-nadir)>=2ng/mL, add uprgflg (unconfirmed PSA progression flag)=1
    - If PSA >=1.25\*nadir and (PSA-nadir)≥ 2ng/mL is confirmed by a second PSA value obtained >=21 days (3 weeks) from the initial increase, add cprgflg (confirmed PSA progression flag)=1

200331

#### PSA response (including PSA50 response)

- If progression is confirmed [sum(uprqflq,cprqflq)=2] output to [PSA progression]
- Else output to [No significant PSA change]
- Step 4. Under Subset II
  - If any visit >=XX days (12 weeks) PSA >= 1.25\*baseline and abs(increase from baseline) >=2ng/mL output to [PSA progression] (no confirmation required).
  - Else output to [No significant PSA change]

#### 13.6.4. Safety

### Adverse Events

#### **AE'S OF Special Interest**

- Hypocalcaemia
- Increase in Creatinine

#### **Duration of AE**

- Calculated as the number of [days] from AE Start Date to AE Stop Date:
  - AE Start Date = Missing
- → Elapse Time = Missing
- AE Stop Date = Missing
- → Elapse Time = Missing

Otherwise

→ Elapsed Time = AE Stop Date – AE Start Date + 1

#### **ECHO/MUGA**

 Change from Baseline for cardiac data, e.g., Left Ventricular Ejection Fraction (LVEF), will be calculated based on the same modality (ECHO or MUGA) throughout the study for each subject. Post-baseline assessments with a different cardiac scan modality will not be used to calculate change from Baseline.

200331

## 13.7. Appendix 7: Reporting Standards for Missing Data

## 13.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as below: • A subject will be considered to have completed the study if the subject dies or otherwise progresses during the study treatment or post-treatment follow-up period. All other subjects will be considered to have withdrawn from the study. |
| | Withdrawn subjects were not replaced in this study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

## 13.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated using a "blank" in subject listing displays. Unless all<br/>data for a specific visit are missing in which case the data is excluded from the<br/>table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 13.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail | |
|---|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. | |
| Adverse<br>Events | <ul> <li>Imputations in the adverse events dataset are used for slotting events to the appropriate study tir periods and for sorting in data listings.</li> <li>Partial dates for AE recorded in the CRF will be imputed using the following conventions:</li> </ul> | ime |
| | Missing start day If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month. Else if study treatment start date is not missing: If month and year of start date = month and year of study treatment start date then If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month. Else set start date = study treatment start date. Else set start date = 1st of month. | |

| Element | Reporting Detail | |
|---|---|---|
| | Missing start day and month Missing stop | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> <li>Last day of the month will be used.</li> </ul> |
| | day Missing stop day and month | No Imputation |
| | Completely<br>missing<br>start/end date | No imputation |
| Concomitant Medications/ Medical | following conve | |
| History/<br>Blood<br>Supportive<br>Products | Missing start day | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing end day | A '28/29/30/31' will be used for the day (dependent on the month and year) |
| | Missing end day and month Completely missing | A '31' will be used for the day and 'Dec' will be used for the month. No imputation |
| New Anti-<br>Cancer | | y-up anti-cancer therapy, radiotherapy (where applicable), and surgical applicable) will be imputed in order to define event and censoring rules for |

| Element | Reporting Detail |
|---|---|
| Therapy/<br>Radiotherap<br>y/<br>Surgical<br>Procedures<br>for Efficacy<br>Evaluation<br>(e.g.,<br>response<br>rate, time to<br>event) | progression-free survival, response rate, or duration of response (i.e. start date for new anticancer therapy). Dates will only be imputed when a month and year are available, but the day is missing. The following rules will be used to impute the date when partial start dates are present on anti-cancer therapy, radiotherapy, and/or surgical procedures dataset[s]: Completely missing start dates will remain missing, with no imputation applied; Partial start dates will be imputed using the following convention: If both month and day are missing, no imputation will be applied; If only day is missing: If the month of partial date is the same as the month of last dosing date, minimum of (last dosing date + 1, last day of the month) will be used for the day; If the month of partial date is the same as the month of last disease assessment and the last disease assessment is PD, minimum of (last date of disease assessment + 1, last day of the month) will be used for the day; If both conditions above are met, the later date will be used for the day; Otherwise, a '01' will be used for the day; |
| | Completely or partial missing end dates will remain missing, with no imputation applied; |
| Treatment end date | If there is more than one study treatment, imputation of missing treatment end date will be applied to all applicable treatments following rules below and treatment end date is the latest treatment end date across all study treatments. For daily oral treatment |
| | <ul> <li>In general, completely missing end dates are not imputed, with the following exceptions for imputation of missing treatment end date at interim analyses.</li> <li>For imputation of missing exposure end date at an interim analysis when subjects are still on treatment, the following conventions will be applied: <ul> <li>If the missing end date is in the last exposure record, the earliest of: the date of the data cut-off, the date of withdrawal from the study, or the death date will be used</li> <li>If the missing end date is not in the last exposure record, treatment start date for the record will be used</li> </ul> </li> <li>The imputed treatment end date will be used to calculate cumulative dose and duration of treatment as specified in Section 13.6.2. For non-continual treatment</li> </ul> |

200331

#### 13.8. Appendix 8: Values of Potential Clinical Importance

#### 13.8.1. Laboratory Values

To identify laboratory values of potential clinical importance, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.0) will be used to assign grades for laboratory parameters including clinical chemistry, haematology, liver function tests, QTc (Bazett's or Fridericia's) values, vital signs (heart rate, blood pressure, temperature) and LVEF.

Reference ranges for all laboratory parameters collected throughout the study are provided by the laboratory. A laboratory value that is outside the reference range is considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Note: a high abnormal or low abnormal laboratory value is not necessarily of clinical concern. The laboratory reference ranges will be provided on the listings of laboratory data. Clinical laboratory test results outside of the reference range will be flagged in the listings.

For laboratory data which are not listed in the NCI CTCAE v4.0, a summary of values outside the normal range will be provided.

#### 13.8.2. ECG and Vital Signs

For ECG and vital signs, the most updated IDSL standard up to the RAP effective date will be followed.

200331

## 13.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

Population PK analysis will be done under a separate RAP and reported outside of the CSR.

200331

# 13.10. Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses

PK/PD analyses will be done under a separate RAP and reported outside of the CSR.

200331

## 13.11. Appendix 11: Abbreviations & Trade Marks

## 13.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALT | Alanine aminotransferase |
| AR | Androgen receptor |
| ATC | Anatomical Therapeutic Chemical |
| AUC | Area under the concentration-time curve |
| AUC(0-t) | Area under the concentration-time curve from zero over the dosing |
| | interval |
| AUC(0-τ) | Area under the concentration-time curve from zero to the last |
| | quantifiable blood or plasma concentration |
| BID | Twice daily |
| BOR | Best Overall Response |
| BP | Blood pressure |
| cfDNA | Circulating-free tumor DNA |
| CI | Confidence Interval |
| CL/F | Oral clearance |
| Cmax | Maximum observed concentration |
| CNV | Copy Number Variant |
| CPMS | Clinical Pharmacology Modeling & Simulation |
| CR | Complete response |
| CSR | Clinical study report |
| CT | Computed tomography |
| CTC | Circulating tumor cells |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DBR | Database Release |
| DBF | Database Freeze |
| DLT | Dose-limiting toxicity |
| DNA | Deoxyribonucleic acid |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| EOS | End of Study |
| EudraCT | European Clinical Trials Database |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Amendments Act |
| FISH | Fluorescent in situ hybridization |
| GSK | GlaxoSmithKline |
| ICH | International Conference on Harmonization |
| IDSL | International Data Standards Library |

| Abbreviation | Description |
|---|---|
| IHC | Immunohistochemistry |
| INDSR | Investigational New Drug Safety Report |
| INR | International Normalized Ratio |
| ka | Absorption rate constant |
| LDH | Lactate dehydrogenase |
| LVEF | Left ventricular ejection fraction |
| M | Mandatory |
| mCRPC | Metastatic castration-resistant prostate cancer |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligrams |
| MHRA | Medicines and Healthcare Products Regulatory Agency |
| mL | Milliliter |
| MRI | Magnetic resonance imaging |
| MTD | Maximum tolerated dose |
| MUGA | Multigated acquisition scan |
| N, n | Number |
| NCI | National Cancer Institute |
| NE NE | Not evaluable |
| O | Optional |
| ORR | Objective Response Rate |
| PCWG2 | Prostate Cancer Working Group 2 |
| PD | |
| ΡΙ3Κβ | Pharmacodynamic or progressive disease |
| PK | Phosphoinositide 3-kinase beta Pharmacokinetic |
| PR | |
| | Partial response |
| PopPK<br>PS | Population Pharmacokinetic Performance Status |
| PSA | |
| PSA50 | Prostate-specific antigen Prostate-specific antigen decrease from baseline >500/ |
| PT | Prostate-specific antigen decrease from baseline ≥50% Prothrombin time |
| PTEN | Phosphatase and tensin homolog |
| PTH | Parathyroid hormone |
| PTT | Partial thromboplastin time |
| Q4wks | Every 4 weeks |
| Q8wks | Every 8 weeks |
| Q12wks | Every 12 weeks |
| QD | Every day |
| QTc | Corrected QT interval |
| QTcB | QT interval corrected by Bazett's formula |
| QTcF | QT interval corrected by Fridericia's formula |
| RAP | Reporting and Analysis Plan |
| RECIST | Response Evaluation Criteria In Solid Tumors |
| RNA | Ribonucleic acid |
| RP2D | Recommended Phase II dose |
| rPFS | Radiological progression free survival |

200331

| Abbreviation | Description |
|--------------|------------------------------------------------------|
| SAC | Statistical Analysis Complete |
| SAE | Serious adverse event(s) |
| SBP | Systolic blood pressure |
| SD | Stable disease or standard deviation |
| SNV | Small Nuclear Variant |
| SRM | Study Reference Manual |
| SRT | Safety Review Team |
| Tmax | Time of occurrence of maximum observed concentration |
| TMF | Trial Master File |
| UPC | Urine protein to creatinine |
| US | United States |
| V/F | Oral volume of distribution |
| Wk(s) | Week(s) |

## 13.11.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| None |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |
200331

#### 13.12. Appendix 12: List of Data Displays

#### 13.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Section | Listings | |
| ICH Listings; | 1 to x | |
| Other Listings | y t | 0 Z |

### 13.12.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays

| Section | Figure | Table | Listing |
|------------------|--------|------------------------|-----------------|
| Study Population | | POP_T1 | |
| Efficacy | | EFF_T1, EFF_T2, EFF_T3 | EFF_L1, EFF_L2 |
| Safety | | | |
| Pharmacokinetic | | | |
| Biomarker | BIO_F1 | | BIO_L1, BIO_L2, |
| | | | BIO_L3 |
| Non-ICH | | | NICH_L1 |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 13.12.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

200331

## 13.12.4. Study Population Tables

| Stud | y Population Tab | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| Subj | ect Disposition | 1 | | 1 | l |
| 1.1. | All Treated<br>Safety | ES8 | Summary of Subject Status and Reason for Study Withdrawal | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | All Treated<br>Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC |
| 1.3. | All Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | EudraCT/Clinical Operations; for all subjects screened; | SAC |
| 1.4. | All Treated<br>Safety | NS1 | Summary of Number of Participant by Country and Site ID | EudraCT/Clinical Operations | SAC |
| 1.5. | All Screened | POP_T1 | Summary of Study Eligibility in Screening | /arenv/arprod/gsk2636771/p3b115717/sac/<br>drivers/t_elig_prescn.sas | SAC |
| Proto | ocol Deviation | 1 | | | L |
| 1.6. | All Treated<br>Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Popu | llation Analysed | 1 | | 1 | |
| 1.7. | All Treated<br>Safety | SP1A | Summary of Study Population | IDSL | SAC |
| Dem | ographic and Bas | seline Characteristi | cs | • | |
| 1.8. | All Treated<br>Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |

| Study | / Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.9. | All Treated<br>Safety | DM11 | Summary of Age Ranges | EudraCT (<18-64, 65-84; >=85); DSUR (<18,18-64, 65-74, >=75) | SAC |
| 1.10. | All Treated<br>Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT; include all races and race details | SAC |
| 1.11. | All Treated<br>Safety | MH1 | Summary of Past Medical Conditions | ICH E3 | SAC |
| 1.12. | All Treated<br>Safety | MH1 | Summary of Current Medical Conditions | ICH E3 | SAC |
| 1.13. | All Treated<br>Safety | CM8 | Summary of Concomitant Medications | ICH E3 | SAC |
| Expo | sure and Treatm | ent Compliance | | <u> </u> | |
| 1.14. | All Treated<br>Safety | EX1 | Summary of Exposure to Study Treatment | ICH E3 | SAC |
| 1.15. | | | | | |
| 1.16. | All Treated<br>Safety | COMP1 | Summary of Overall Compliance Based on Exposure | | SAC |
| Disea | se Characteristi | cs | | ' | - |
| 1.17. | All Treated<br>Safety | DC1 | Summary of Disease Characteristics at Initial Diagnosis | ICH E3; See Table 1.4 from /arenv/arprod/gsk2636771/mid200331/ | SAC |
| | Salety | | | dsur_2018_01/drivers/t_dischar_init.sas | |
| 1.18. | All Treated<br>Safety | DC2 | Summary of Disease Characteristics at Screening | See Table 1.5 from /arenv/arprod/<br>gsk2636771/mid200331/ | SAC |

| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| | | | | dsur_2018_01/drivers/ | |
| | | | | t_dischar_scr.sas add | |
| | | | | Time on Enza prior study, | |
| 1.19. | All Treated<br>Safety | LA1 | Summary of Disease Burden at Baseline | ICH E3 | SAC |
| Anti-0 | Cancer Therapy | • | | | |
| 1.20. | All Treated<br>Safety | AC2 | Summary of Prior Anti-Cancer Therapy | IDSL; add "Enzalutamide received prior to chemotherapy", "Enzalutamide received following chemotherapy" | SAC |
| 1.21. | All Treated<br>Safety | CM1 | Summary of Pre-Treatment Dictionary Coded Anti-Cancer Therapy | IDSL | SAC |
| 1.22. | All Treated<br>Safety | CM1 | Summary of Post-Treatment Dictionary Coded Anti-Cancer Therapy | IDSL | SAC |
| 1.23. | All Treated<br>Safety | AC3 | Summary of Number of Prior Anti-Cancer Therapy Regimens | IDSL; include Biologic, chemotherapy, hormonal, immunotherapy, radioactive therapy, and small molecule targeted therapy along with radiotherapy and surgery | SAC |
| 1.24. | All Treated | AC4 | Summary of Best Response to Prior Enzalutamide Therapy | | SAC |
| 1.25. | All Treated<br>Safety | AC4 | Summary of the Most Recent Best Response to Prior Anti-<br>Cancer Therapies | IDSL; By therapies | SAC |
| 1.26. | All Treated<br>Safety | FAC1 | Summary of Post-Treatment Anti-Cancer Therapy | IDSL; include Biologic, chemotherapy, hormonal, immunotherapy, radioactive therapy, and small molecule targeted therapy along with radiotherapy and | SAC |

| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| | | | | surgery | |
| Surg | ical and Medical | Procedures | | · | 1 |
| 1.27. | All Treated<br>Safety | OSP1 | Summary of Prior Cancer-Related Surgical Procedures | IDSL, include follow-up surgeries separately if present | SAC |
| Subs | stance Use | | | , | 1 |
| 1.28. | All Treated | SU1 | Summary of Substance Use | IDSL, include Smoking history and alcohol | SAC |

#### 200331

## 13.12.5. Efficacy Tables

| Effica | cy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverabl<br>e [Priority] |
| 2.1. | Modified All<br>Treated Clinical<br>Activity | EFF_T1 | Summary of Confirmed and Unconfirmed Non-PD Response Rate at 12 Weeks (PCWG2 Criteria) | Include 95% exact confidence interval | SAC |
| 2.2. | All Treated<br>Clinical Activity | RE1a | Summary of Investigator-Assessed Best Response (RECIST 1.1 Criteria) (Confirmed) for Subjects with Target Lesion and/or Non-Target Lesion at Baseline | Including response <u>without</u> <u>confirmation</u> ; (see Table 2.006 present_2016_1 reporting effort) | SAC |
| 2.3. | All Treated<br>Clinical Activity | RE1a | Summary of Investigator-Assessed Best Response (RECIST 1.1 Criteria) (Unconfirmed) for Subjects with Target Lesion and/or Non-Target Lesion at Baseline | Including response with confirmation; (see Table 2.007 from present_2016_1 reporting effort) | SAC |
| 2.4. | All Treated<br>Clinical Activity | EFF_T2 | Summary of PSA50 Response for All Subjects (Confirmed) | Including response with confirmation (see Table 2.008 from present_2016_1 reporting effort), provide overall results and results stratified by measurable vs. non-measurable disease at baseline | SAC |
| 2.5. | All Treated<br>Clinical Activity | EFF_T2 | Summary of PSA50 Response for All Subjects (Unconfirmed) | Including response without confirmation (see Table 2.009 from present_2016_1 reporting effort), provide overall results and results stratified by measurable vs. non-measurable disease at baseline | SAC |
| 2.6. | All Treated<br>Clinical Activity | TTE1 | Summary of Time to PSA progression (PCWG2 criteria) | Add footnote indicating 400 mg cohort not summarized individually due to small sample size (n=2) | SAC |
| 2.7. | All Treated<br>Clinical Activity | TTE1 | Summary of Time to radiological progression (PCWG2 criteria) | Add footnote indicating 400 mg cohort not summarized individually due to small sample size (n=2) | SAC |
| 2.8. | All Treated<br>Clinical Activity | TTE1 | Summary of Investigator-Assessed Radiological Progression-Free Survival (PCWG2 Criteria) | Add footnote indicating 400 mg cohort not summarized individually due to small sample size (n=2) | SAC |

200331

## 13.12.6. Efficacy Figures

| Efficacy: | Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverabl<br>e [Priority] |
| 2.1 | All Treated<br>Clinical<br>Activity | | Waterfall Plot of Maximum Reduction in PSA Values by Dose | arenv/arprod/gsk2636771/mid2003<br>31/present_2018_01/drivers/f_wate<br>r_psa.sas | SAC |
| 2.2 | All Treated<br>Clinical<br>Activity | OLB12B | Mean Change (95% CI) Change from Baseline in PSA by Time and Treatment | | SAC |
| 2.3 | All Treated<br>Clinical<br>Activity | | Spider Plot of Percent Change from Baseline in PSA values by Dose | arenv/arprod/gsk2636771/mid2003<br>31/present_2018_01/drivers/f_spid<br>er_psa_1.sas | SAC |
| 2.4 | All Treated<br>Clinical<br>Activity | | Waterfall Plot of Maximum Reduction in Target Lesion Diameter by Dose | arenv/arprod/gsk2636771/mid2003<br>31/present_2018_01/drivers/f_delta<br>_p1.sas | SAC |
| 2.5 | All Treated<br>Clinical<br>Activity | | Spider Plot of Percent Change from Baseline in Target Lesion<br>Diameter by Dose | arenv/arprod/gsk2636771/mid2003<br>31/present_2018_01/drivers/f_spid<br>er_nmc_2.sas | SAC |
| 2.6 | All Treated<br>Clinical<br>Activity | OEX12 | Swimming Lane Plot of Duration of Study Treatment by Dose | One panel for each cohort; add labels of PR, PSA PD, Radiological PD, clinical PD, DLT, AEs leading to dose reduction/interruption etc. | SAC |
| 2.7 | All Treated<br>Clinical<br>Activity | TTE10 | Graph of Kaplan Meier Investigator-Assessed Radiological Progression-Free Survival Curves by dose | Do not summarize results for the 400 mg cohort | SAC |

200331

| Efficacy: | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverabl<br>e [Priority] |
| 2.8 | All Treated<br>Clinical<br>Activity | TTE10 | Graph of Kaplan Meier Investigator-Assessed Radiological Progression-Free Survival Curves (overall) | 400 mg included in overall summary | SAC |
| 2.9 | All Treated<br>Clinical<br>Activity | TTE10 | Graph of Kaplan Meier Curves for Time to PSA Progression by dose | Do not summarize results for the 400 mg cohort | SAC |
| 2.10 | All Treated<br>Clinical<br>Activity | TTE10 | Graph of Kaplan Meier Curves for Time to PSA Progression (overall) | 400 mg included in overall summary | SAC |
| 2.11 | All Treated<br>Clinical<br>Activity | TTE10 | Graph of Kaplan Meier Curves for Time to Radiological Progression by dose | Do not summarize results for the 400 mg cohort | SAC |
| 2.12 | All Treated<br>Clinical<br>Activity | TTE10 | Graph of Kaplan Meier Curves for Time to Radiological Progression (overall) | 400 mg included in overall summary | SAC |

# 13.12.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Adverse Events (AEs) | | | | |
| 3.1. | All Treated<br>Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.2. | All Treated<br>Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | ICH E3 | SAC |
| 3.3. | All Treated<br>Safety | AE3 | Summary of Common (>=5%) Grade 2-4 Adverse Events by Overall Frequency | ICH E3 | SAC |
| 3.4. | All Treated<br>Safety | AE3 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade | ICH E3 | SAC |
| 3.5. | All Treated<br>Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term and Maximum Grade | FDAAA, EudraCT | SAC |
| 3.6. | All Treated<br>Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4 Adverse Events by Overall Frequency | ICH E3 | SAC |
| 3.7. | All Treated<br>Safety | OAE07 | Summary of All Adverse Events by Maximum Grade | | SAC |
| 3.8. | All Treated<br>Safety | OAE07 | Summary of Adverse Events Related to Study Treatment by Maximum Grade | | SAC |
| 3.9. | All Treated<br>Safety | AE3 | Summary of Adverse Events Leading to Dose Reductions | By preferred term | SAC |
| 3.10. | All Treated<br>Safety | AE3 | Summary of Adverse Events Leading to Dose Escalations | By preferred term | SAC |
| 3.11. | All Treated<br>Safety | AE3 | Summary of Adverse Events Leading to Dose Interruptions | By preferred term | SAC |
| Adverse | Events of Specia | al Interest | | | • |
| 3.12. | All Treated<br>Safety | ESI1 | Summary of Characteristics of Hypocalcaemia | | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.13. | All Treated<br>Safety | ESI2a | Summary of Onset and Duration of the First Occurrence of<br>Hypocalcaemia | | SAC |
| 3.14. | All Treated<br>Safety | OAE01 | Summary of Hypocalcaemia by Maximum Grade | by AESI and preferred term | SAC |
| 3.15. | All Treated<br>Safety | AE17 | Summary of Exposure Adjusted Incidence Rate for Hypocalcaemia by Maximum Grade | | SAC |
| 3.16. | All Treated<br>Safety | ESI1 | Summary of Characteristics of Increase in Creatinine | | SAC |
| 3.17. | All Treated<br>Safety | ESI2a | Summary of Onset and Duration of the First Occurrence of Increase in Creatinine | | SAC |
| 3.18. | All Treated<br>Safety | OAE01 | Summary of Increase in Creatinine by Maximum Grade | by AESI and preferred term | SAC |
| 3.19. | All Treated<br>Safety | AE17 | Summary of Exposure Adjusted Incidence Rate for Increase in Creatinine by Maximum Grade | | SAC |
| Serious | and Other Signifi | cant Adverse I | Events | | |
| 3.20. | All Treated<br>Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC |
| 3.21. | All Treated<br>Safety | AE3 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by Preferred Term | | SAC |
| 3.22. | All Treated<br>Safety | AE3 | Summary of Serious Adverse Events by Maximum Grade | By preferred term | SAC |
| 3.23. | All Treated<br>Safety | AE3 | Summary of Drug Related Serious Adverse Events by Maximum Grade | By preferred term | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.24. | All Treated<br>Safety | AE3 | Summary of Fatal Adverse Events | If there are < 5 fatal AEs, only provide listing. | SAC |
| 3.25. | All Treated<br>Safety | AE3 | Summary of Drug Related Fatal Adverse Events | If there are < 5 fatal AEs, only provide listing. | SAC |
| 3.26. | All Treated<br>Safety | AE3 | Summary of Non-Serious Drug-Related Adverse Events by Overall Frequency | | SAC |
| 3.27. | All Treated<br>Safety | AE3 | Summary of Serious Drug-Related Adverse Events by Overall Frequency | | SAC |
| Deaths | | | | | |
| 3.28. | All Treated<br>Safety | DTH1A | Summary of Deaths | IDSL; report time to death from last dose in weeks | SAC |
| 3.29. | All Treated<br>Safety | AE5 | Summary of Cardiovascular Events by maximum Grade | See Section 8.6.1 for details. | SAC |
| Labora | tory: Chemistry | | | | |
| 3.30. | All Treated<br>Safety | LB1 | Summary of Chemistry Changes from Baseline | ICH E3; include PSA, serum testosterone, and PTH, ionized calcium, vitamin D (total D, D1, D2, and D3), Serum Bone Markers (osteocalcin, Bone Specific Alk Phos, Serum N-telopeptide) | SAC |
| 3.31. | All Treated<br>Safety | LB1 | Summary of Percent Changes in Chemistry from Baseline | include PSA, serum testosterone, and PTH, ionized calcium, vitamin D (total D, D1, D2, and D3), Serum Bone Markers (osteocalcin, Bone Specific Alk Phos, Serum N-telopeptide) | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.32. | All Treated<br>Safety | OLB9C | Summary of Worst Case Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3; by visit summary rows are not needed | SAC |
| 3.33. | All Treated<br>Safety | OLB11B | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | SAC |
| Laborat | tory: Haematology | у | | | |
| 3.34. | All Treated<br>Safety | LB1 | Summary of Haematology Changes from Baseline | ICH E3; include PT, PTT, and INR | SAC |
| 3.35. | All Treated<br>Safety | LB1 | Summary of Percent Changes in Haematology from Baseline | include PT, PTT, and INR | SAC |
| 3.36. | All Treated<br>Safety | OLB9C | Summary of Worst Case Haematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3; by visit summary rows are not needed | SAC |
| 3.37. | All Treated<br>Safety | OLB11B | Summary of Worst Case Haematology Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | SAC |
| Laborat | tory: Urinalysis | | | | |
| 3.38. | All Treated<br>Safety | LB1 | Summary of Urine Concentration Changes from Baseline | ICH E3; include Urine Bone Marker (Urine C-telopeptide), | SAC |
| 3.39. | All Treated<br>Safety | LB1 | Summary of Percent Changes in Urine Concentration from Baseline | include Urine Bone Marker (Urine C-telopeptide), | SAC |
| 3.40. | All Treated<br>Safety | OUR1B | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | ICH E3 | |
| Laborat | tory: Hepatobiliar | y (Liver) | | | |
| 3.41. | All Treated<br>Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.42. | All Treated<br>Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC |
| ECG | | | | | |
| 3.43. | All Treated<br>Safety | EG1 | Summary of ECG Findings | IDSL | SAC |
| 3.44. | All Treated<br>Safety | OECG1B | Summary of Maximum Fridericia's QTc Values Post-Baseline Relative to Baseline by Category | IDSL | SAC |
| 3.45. | All Treated<br>Safety | EG2 | Summary of Change from Baseline in ECG values by Visit | IDSL | SAC |
| 3.46. | All Treated<br>Safety | OECG2B | Summary of Maximum Increase in Fridericia's QTc Values Post-<br>Baseline Relative to Baseline by Category | IDSL | SAC |
| Vital Si | gns | • | | | • |
| 3.47. | All Treated<br>Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC |
| 3.48. | All Treated<br>Safety | OVT2B | Summary of Worst Case Vital Signs Results by Maximum Grade Increase Post-Baseline Relative to Baseline | IDSL | SAC |
| 3.49. | All Treated<br>Safety | OVTB | Summary of Worst Case Vital Signs Results Relative to Normal Range Post-Baseline Relative to Baseline | IDSL | SAC |
| LVEF | | | | | • |
| 3.50. | All Treated<br>Safety | OLVEF1A | Summary of Left Ventricular Ejection Fraction (%) Absolute Change from Baseline | IDSL; Add "(%) Absolute" in title; remove column "LVEF (%)" | SAC |
| Dose M | odifications | | | | |
| 3.51. | All Treated<br>Safety | ODMOD1 | Summary of Dose Reductions of GSK2636771 | ICH E3 | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.52. | All Treated<br>Safety | ODMOD1 | Summary of Dose Escalations of GSK2636771 | ICH E3 | SAC |
| 3.53. | All Treated<br>Safety | ODMOD2 | Summary of Dose Interruptions of GSK2636771 | ICH E3 | SAC |
| 3.54. | All Treated<br>Safety | ODMOD1 | Summary of Dose Reductions of Enzalutamide | ICH E3 | SAC |
| 3.55. | All Treated<br>Safety | ODMOD1 | Summary of Dose Escalations of Enzalutamide | ICH E3 | SAC |
| 3.56. | All Treated<br>Safety | ODMOD2 | Summary of Dose Interruptions of Enzalutamide | ICH E3 | SAC |
| Dose Li | imiting Toxicity (D | LT) | | | |
| 3.57. | All Treated<br>Safety | DL1 | Summary of Dose-Limiting Toxicities during the Determinative Period | ICH E3 | SAC |
| Perform | nance Status | | | | · |
| 3.58. | All Treated<br>Safety | PS1A | Summary of ECOG Performance Status | ICH E3 | SAC |
| 3.59. | All Treated<br>Safety | PS4A | Summary of Change in ECOG Performance Status from Baseline | | SAC |

200331

## 13.12.8. Safety Figures

| Safety: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Events | | | | |
| 3.1. | All Treated<br>Safety | AE10 | Plot of Common (>=5%) Adverse Events | IDSL | SAC |
| Laborato | ory | | | | |
| 3.2. | All Treated<br>Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin | IDSL | SAC |
| 3.3. | All Treated<br>Safety | LB11 | Figure of LFT Patient Profiles for Possible Hy's Law Subjects by Dose | If there are subjects with liver events | SAC |
| 3.4. | All Treated<br>Safety | LB7 | Summary of change from Baseline in Calcium values by Dose (Hypocalcaemia, hypophosphatemia, creatinine increase) | | SAC |
| ECG | | • | | <u>.</u> | |
| 3.5. | All Treated<br>Safety | OECG4 | Fridericia's QTc Shifts from Baseline to Worst-case Post Baseline | IDSL | SAC |

200331

### 13.12.9. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| PK Cor | ncentration | | | | |
| 4.1. | PK concentration | PK01 | Summary of GSK2636771 (in the presence of enzalutamide) Plasma Pharmacokinetic Concentration-Time Data by dose | IDSL | SAC |
| 4.2. | PK concentration | PK01 | Summary of Enzalutamide Plasma Pharmacokinetic Concentration-Time Data by Dose (with and without GSK2636771) | IDSL | SAC |
| 4.3. | PK concentration | PK01 | Summary of N-desmethyl enzalutamide Plasma Pharmacokinetic Concentration-Time Data by Dose (with and without GSK2636771) | IDSL | SAC |

200331

## 13.12.10. Pharmacokinetic Figures

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK | | | | | |
| 4.1. | PK concentration | PK16a | Individual GSK2636771 (in the presence of enzalutamide) Concentration-Time Plots (Linear and Semi-log) - Dose Escalation Phase only | IDSL | SAC |
| 4.2. | PK concentration | PK17 | Mean GSK2636771 (in the presence of enzalutamide) Concentration-Time Plots (Linear and Semi-log) by Dose - Dose Escalation Phase only | IDSL | SAC |
| 4.3. | PK concentration | PK18 | Median GSK2636771 (in the presence of enzalutamide) Concentration-Time Plots (Linear and Semi-log) by Dose - Dose Escalation Phase only | IDSL | SAC |
| 4.4. | PK concentration | PK16a | Individual Enzalutamide Concentration-Time Plots (Linear and Semi-log) - Dose Escalation Phase only (with and without GSK2636771) | IDSL | SAC |
| 4.5. | PK concentration | PK17 | Mean Enzalutamide Concentration-Time Plots (Linear and Semilog) by Dose- Dose Escalation Phase only (with and without GSK2636771) | IDSL | SAC |
| 4.6. | PK concentration | PK18 | Median Enzalutamide Concentration-Time Plots (Linear and Semi-log) by Dose- Dose Escalation Phase only (with and without GSK2636771) | IDSL | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.7. | PK concentration | PK16a | Individual N-desmethyl enzalutamide Concentration-Time Plots (Linear and Semi-log) - Dose Escalation Phase only (with and without GSK2636771) | IDSL | SAC |
| 4.8. | PK concentration | PK17 | Mean N-desmethyl enzalutamide Concentration-Time Plots (Linear and Semi-log) by Dose- Dose Escalation Phase only (with and without GSK2636771) | IDSL | SAC |
| 4.9. | PK concentration | PK18 | Median N-desmethyl enzalutamide Concentration-Time Plots (Linear and Semi-log) by Dose- Dose Escalation Phase only (with and without GSK2636771) | IDSL | SAC |
| 4.10. | PK Concentration | PK19 | Mean enzalutamide and GSK2636771 (by dose) Concentration-<br>Time Plots (with and without GSK2636771) | Plot GSK2636771 concentrations by dose | SAC |
| 4.11. | PK Concentration | PK19 | Mean N-desmethyl enzalutamide and GSK2636771 (by dose)<br>Concentration-Time Plots (with and without GSK2636771) | Plot GSK2636771 concentrations by dose | SAC |

200331

### 13.12.11. Biomarker Tables

| Biomarl | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.1 | Biomarker | BIO_T1 | Summary of Conversion (>5 cells/mL dropping to ≤5 cells/mL) from Baseline in CTCs by Visit | | SAC |
| 5.2 | All Screened | BIO_T2 | Summary of Frequency of PTEN Loss (H-Score ≤ 30) at Screening | | SAC |
| 5.3 | Biomarker | BIO_T3 | Categorization of PTEN loss by Sequencing (homozygous vs heterozygous) | | SAC |

## 13.12.12. Biomarker Figures

| Biomark | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.1 | Biomarker | BIO_F1 | Heatmap Display of 2 or More Gene Alterations by Subject | | SAC |

200331

## 13.12.13. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | All Enrolled | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | All Treated Safety | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | All Treated Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| 4. | All Treated Safety | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 5. | All Treated Safety | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 6. | All Treated Safety | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | |
| 7. | All Treated Safety | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | SAC |
| Demog | raphic and Baseline Ch | naracteristics | | | |
| 8. | All Treated Safety | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 9. | All Treated Safety | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | nd Concomitant Medica | ations | | | |
| 10. | All Treated Safety | CP_CM3 | Listing of Concomitant Medications | IDSL | SAC |
| Expos | ure and Treatment Com | pliance | 1 | | <u></u> |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 11. | All Treated Safety | OEX3A | Listing of Exposure to Enzalutamide | ICH E3 | SAC |
| 12. | All Treated Safety | OEX3A | Listing of Exposure to GSK2636771 | | SAC |
| 13. | All Treated Safety | COMP2 | Listing of Study Treatment Compliance | | SAC |
| 14. | All Treated Safety | ODMOD10a | Listing of Dose Reductions | | SAC |
| 15. | All Treated Safety | ODMOD10a | Listing of Dose Escalations | | SAC |
| 16. | All Treated Safety | ODMOD11a | Listing of Dose Interruptions | | SAC |
| Respoi | nse | | | | |
| 17. | Modified All Treated<br>Clinical Activity | EFF_L1 | Listing of Overall Unconfirmed Response at Week 12 | List all data used for Table 2.1 by cohort and subject – see Listing 2.010 from reporting effort present_2016_1 | SAC |
| 18. | Modified All Treated<br>Clinical Activity | EFF_L1 | Listing of Overall Confirmed Response at Week 12 | List all data used for Table 2.1 by cohort and subject – see Listing 2.010 from reporting effort present_2016_1 | SAC |
| 19. | All Treated Clinical<br>Activity | LA2 | Listing of Investigator Assessed Target Lesion<br>Assessments (RECIST 1.1 Criteria) | | SAC |
| 20. | All Treated Clinical<br>Activity | LA3 | Listing of Investigator-Assessed Non-Target Lesion Assessments (RECIST 1.1 Criteria) | | SAC |
| 21. | All Treated Clinical<br>Activity | LA4 | Listing of Investigator -Assessed New Lesions (RECIST 1.1 Criteria) | | SAC |
| 22. | All Treated Clinical<br>Activity | RE5 | Listing of Investigator -Assessed Tumour Responses(RECIST1.1 Criteria) | Include with and without confirmation in same listing | SAC |
| 23. | All Treated Clinical<br>Activity | OLB7 | Listing of Subject PSA Value by Visit/Week | | SAC |
| 24. | All Treated Clinical<br>Activity | LA2 | Listing of Subject Bone Scan Results by Visit/Week | Use lesion dataset where lsorgcd=BE | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 25. | All Treated Clinical<br>Activity | TTE9 | Listing of Time to PSA Progression | | SAC |
| 26. | All Treated Clinical<br>Activity | TTE9 | Listing of Time to Radiological Progression | | SAC |
| 27. | All Treated Clinical<br>Activity | TTE9 | Listing of Radiographic Progression-Free Survival | | SAC |
| Advers | se Events | | | | |
| 28. | All Treated Safety | AE8 | Listing of All Adverse Events | ICH E3 | SAC |
| 29. | All Treated Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 30. | All Treated Safety | AE2 | Listing of Relationship Between System Organ Class, Preferred Terms and Verbatim Text | IDSL | SAC |
| Seriou | s and Other Significant | Adverse Events | | | |
| 31. | All Treated Safety | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | SAC |
| 32. | All Treated Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC |
| 33. | All Treated Safety | AE14 | Listing of Reasons for Considering as a Serious<br>Adverse Event | ICH E3 | SAC |
| 34. | All Treated Safety | AE8 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| 35. | All Treated Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study | ICH E3 | SAC |
| Dose L | imiting Toxicities | | | | • |
| 36. | All Treated Safety | DL3 | Listing of Dose-Limiting Toxicities (DLTs) During the Determinative Period | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Deaths | | | | | |
| 37. | All Treated Safety | DTH3 | Listing of Deaths | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | | |
| 38. | All Treated Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC |
| 39. | All Treated Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC |
| All Lab | oratory | | | | |
| 40. | All Treated Safety | LB5A | Listing of All Laboratory Data for Participants with Any Value Outside Normal Range | ICH E3; include PSA, serum testosterone, parathyroid hormone, PT, PTT, INR | SAC |
| 41. | All Treated Safety | LB5A | Listing of All Bone Biomarker Laboratory Data | Include ionized calcium, vitamin D (total D, D1, D2, and D3), Urine Bone Marker (Urine C-telopeptide), Serum Bone Markers (osteocalcin, Bone Specific Alk Phos, Serum N-telopeptide) | SAC |
| 42. | All Treated Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| 43. | All Treated Safety | UR2A | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| ECG | | | | | |
| 44. | All Treated Safety | EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 45. | All Treated Safety | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 46. | All Treated Safety | OECG5A | Listing of Fridericia's QTc Values of Potential Clinical Importance | | SAC |
| Vital Signs | | | | | |
| 47. | All Treated Safety | OVT7A | Listing of Vital Signs with Values of Potential Clinical Importance | | SAC |
| Performance Status | | | | | |
| 48. | All Treated Safety | PS5A | Listing of Performance Status | | SAC |

200331

# 13.12.14. Non-ICH Listings

| Non-I | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Disea | se Characteristic | CS | | | |
| 49. | All Treated<br>Safety | DC3 | Listing of Disease Characteristics at Initial Diagnosis | | SAC |
| 50. | All Treated<br>Safety | DC4 | Listing of Disease Characteristics at Screening | | SAC |
| 51. | All Treated<br>Safety | MD2 | Listing of Metastatic Disease at Screening | | SAC |
| 52. | All Treated<br>Safety | MH2 | Listing of Current and Past Medical Conditions | Only required is conditions are not MedDRA coded | SAC |
| Anti-C | ancer Therapy | | | | |
| 53. | All Treated<br>Safety | AC6 | Listing of Prior Anti-Cancer Therapy | | SAC |
| 54. | All Treated<br>Safety | AC7 | Listing of Prior Anti-Cancer Radiotherapy | | SAC |
| 55. | All Treated<br>Safety | AC6 | Listing of Follow-up Anti-Cancer Therapy | | SAC |
| 56. | All Treated<br>Safety | AC7 | Listing of Follow-up Anti-Cancer Radiotherapy | | SAC |
| Surgio | cal Procedures | 1 | | | |
| 57. | All Treated<br>Safety | OSP3 | Listing of Prior/Post-Treatment Cancer Related Surgical Procedures | | SAC |

| Non-l | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subst | Substance Use | | | | |
| 58. | All Treated<br>Safety | SU2 | Listing of Substance Use | | SAC |
| Respo | onses | | | | |
| 59. | All Treated<br>Clinical<br>Activity | RE6 | Listing of Subjects with Progressive Disease Based on Clinical Assessment | | SAC |
| LVEF | | | | | |
| 60. | All Treated<br>Safety | OLVEF2A | Listing of Left Ventricular Ejection Fraction Results | Option | SAC |
| PK | | | | | |
| 61. | PK<br>Concentration | PK07 | Listing of GSK2636771 (in the presence of enzalutamide) Pharmacokinetic Concentration-Time Data by Dose | IDSL | SAC |
| 62. | PK<br>Concentration | PK07 | Listing of Enzalutamide Pharmacokinetic Concentration-Time Data by Dose | IDSL | SAC |
| 63. | PK<br>Concentration | PK07 | Listing of N-desmethyl enzalutamide Pharmacokinetic Concentration-<br>Time Data by Dose | IDSL | SAC |
| Other | | | | | |
| 64. | All Treated<br>Safety | NICH_L1 | Listing of Subjects Received Blood Product or Blood Supportive Care | Including all data in BLDPROD dataset | SAC |
| 65. | All Treated<br>Safety | | Listing of Circulating Tumour Cells (CTC) Concentrations | arenv/arprod/gsk2636771/p3b115717/sac/<br>drivers/t_ctc.sas; add column indicating<br>whether there have been conversion to <<br>5 cells/7.5mL from week 1. | SAC |

| Non-I | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 66. | All Treated<br>Safety | OLIVER5 | Listing of Liver Chemistry Assessments for Subjects with Liver Signal/Events | | SAC |
| 67. | All Treated<br>Safety | PREG1a | Listing of Pregnancies | update for partners who became pregnant | SAC |

200331

## 13.13. Appendix 13: Example Mock Shells for Data Displays

Data Display Specification will be made available on request